

# Non-Interventional Study Protocol 747-404/405 OBETICHOLIC ACID (OCA)

# Replicate Studies Evaluating the Effectiveness of Obeticholic Acid on <u>He</u>patic <u>Real-World Outcomes</u> in Patients with <u>Primary Biliary Cholangitis</u> (HEROES PBC)

Version 1.0: 24 January 2022

ClinicalTrials.gov Identifier: NCT05292872

# Sponsor

Intercept Pharmaceuticals, Inc. 305 Madison Avenue Morristown, New Jersey 07960

USA

**TEL:** +1 858 652 6800

FAX: +1 858 558 5961

#### CONFIDENTIAL

The information contained herein is the property of Intercept Pharmaceuticals, Inc. and may not be reproduced, published, or disclosed to others without written authorization of Intercept Pharmaceuticals, Inc.

# SPONSOR'S APPROVAL OF THE PROTOCOL

# 

, MD Date

Intercept Pharmaceuticals, Inc.

─8E73D4F5994B4BC9B7F001BB15A29732

# **INVESTIGATOR'S AGREEMENT**

I have received and read the current version of the Investigator's Brochure (IB) for obeticholic acid (OCA) and this Protocol 747-404/405. Having fully considered all the information available, I agree that it is ethically justifiable to conduct this study according to this protocol.

I understand that all information concerning OCA supplied to me by the Sponsor, Intercept Pharmaceuticals, Inc., and/or its agents in connection with this study and not previously published is confidential information. This includes the IB, study protocol and any other preclinical and clinical data provided by the Sponsor.

I understand that no data are to be made public or published without prior knowledge and written approval by the Sponsor.

By my signature below, I hereby attest that I have read, understood and agreed to abide by all the conditions, instructions and restrictions contained in Protocol 747-404/405 and in accordance with the elements of Good Clinical Practice (CPMP/ICH/135/95) and the Declaration of Helsinki relevant to observational research, and all regulatory requirements for protection of human subjects in studies and privacy requirements for the protection of individual and company data.

I acknowledge that the Sponsor of the study has the right to discontinue the study at any time.

| Investigator's Name (Printed) | |
|-------------------------------|------|
| Investigator's Signature | Date |

# STUDY PERSONNEL CONTACT INFORMATION

# **Sponsor Contact Information**

Primary Contact: PhD

Global Medical Affairs

Intercept Pharmaceuticals Inc. (Intercept)

Telephone:

Email:

# **SAE Reporting Information**

SAE Fax: +1 800 497 8521

ISAE Email: sae@interceptpharma.com

# Or if Not Available:

Contact: MD

Scientific Affairs

Intercept

Telephone:

Email:

# 1. SYNOPSIS

#### Name of Sponsor/Company:

Intercept Pharmaceuticals, Inc.

# Name of Investigational Product:

Obeticholic Acid

#### Name of Active Ingredient:

Obeticholic acid (OCA); 6α-ethyl-chenodeoxycholic acid; (6-ECDCA); INT-747; DSP-1747

# Title of Study:

Replicate Studies Evaluating the Effectiveness of Obeticholic Acid on Hepatic Real-World Outcomes in Patients with Primary Biliary Cholangitis (HEROES PBC)

# **Investigators and/or Study Center(s):**

Alexander Breskin (Target, University of North Carolina - Chapel Hill)

M. Alan Brookhart (Target, Duke University)

Michael Fried (Target)

Bettina Hansen (University Health Network)

Gideon Hirschfield (University Health Network)

John Seeger (Optum)

David Thompson (Syneos Health)

Rajeshwari Punekar (Syneos Health)

#### Studied Period (years):

Estimated initial patient inclusion date 01 Jun 2015

Estimated date last patient observation: 31 Dec 2021

#### **Phase of Development:**

Phase 4

#### **Objectives:**

#### Primary Objective

To evaluate the effect of OCA treatment on time to the first occurrence of the composite endpoint of all-cause death, liver transplant, or hospitalization for hepatic decompensation in PBC patients in 2 data sources: Global PBC registry and Komodo Health claims database.

#### **Exploratory Objectives:**

To evaluate the effect of OCA treatment on time to the first occurrence of individual components of the composite endpoint (outlined below):

- All-cause death
- Liver transplant
- Hospitalization for hepatic decompensation based on the first occurrence of:
  - Variceal bleed
  - o Ascites (including hepatic hydrothorax and spontaneous bacterial peritonitis)
  - Hepatic encephalopathy

#### Methodology:

These are replicate, observational, retrospective cohort studies of patients with PBC who failed ursodeoxycholic acid (UDCA) treatment using 2 real-world data sources: the Global PBC registry (Study 747-404) and the Komodo Health United States (US) claims database (Study 747-405). All analyses will be conducted separately by data source (ie, not pooled). The primary endpoint is time to first occurrence of all-cause death, liver transplant, or hospitalization for hepatic decompensation. The analytic approach is a nested target trial emulation design.

The Komodo Health database contains administrative claims from >350 US payers, including commercial (63%); Medicaid (23%); Medicare (10%); dual eligible (<1%); and other (2%). Data are tokenized to allow for patient tracking across payers. Komodo Health claims will be linked through Datavant tokenization to Quest Diagnostics and LabCorp laboratory data, the US National Death Index (NDI), and the Organ Transplant Network (OPTN) transplant registry for additional information and outcome verification. The database contains >100,000 patients with a PBC diagnostic code. The Global PBC registry includes >5,000 patients with PBC recruited from 17 liver centers across 8 countries in Europe and North America. It utilizes the CASTOR trial platform for electronic case report form (eCRF) collection of medical history, clinical events, and laboratory and treatment data.

All patients who meet diagnostic criteria for PBC in each database between 01 Jun 2015 and 31 Dec 2021 and who meet all eligibility criteria will be considered for these studies. The OCA treatment evaluation period will be from 01 Jun 2016 (based on first country approval by Food and Drug Administration on 27 May 2016). The Komodo Health database is US-specific and the Global PBC registry includes the US and multiple other countries with later approval dates. The Sponsor has applied the date of first global approval of 01 Jun 2016 for both studies. The first date of prescription of OCA after inadequate UDCA response (ALP>upper limit of normal [ULN] and/or total bilirubin [TB]>ULN after >270 days of treatment) or UDCA intolerance (discontinued UDCA after <90 days despite ALP>ULN and/or TB>ULN) will be defined as the index date for OCA-treated PBC patients. The dates of evidence of inadequate UDCA response or UDCA intolerance during which OCA is not utilized will be used as an index date for the non–OCA-treated comparator group.

Each time a patient meets the UDCA inadequate response/intolerance definition or the definition of OCA initiation, in addition to all other eligibility criteria, they will contribute an index to the study. Therefore, patients may contribute multiple control indices, and may contribute control indices before OCA initiation, but can contribute only one OCA initiation index. The non–OCA-treated patient indices will be weighted to have the same baseline covariate distribution as the OCA-treated patients at the time of OCA initiation, thus allowing for the estimation of the effect of treatment in the treated patients. The pre-index period is defined as 12 months prior to the index date, and follow-up is until the first occurrence of any component of the composite endpoint. Patients will be censored at dropout/disenrollment from the database, discontinuation of OCA (+90 days), initiation of fenofibrate or bezafibrate, initiation of OCA (for the non–OCA-treated patient -indices), unapproved OCA dose (>10 mg once daily [QD]) for those treated with OCA, or the end of the study period (31 Dec 2021), whichever comes first.

#### Schematic Diagram Studies 747-404/405:



#### **Number of Patients (planned):**

<u>Komodo Health</u>: In the current Komodo Health database, there are 395 patients who meet all of the following criteria for the OCA treatment group:

- Meet PBC claims diagnostic criteria (1 inpatient or 2 outpatient claims)
- Have evidence of UDCA failure
- Have initiated OCA treatment

There are 5916 patients who meet all of the following criteria for the control group (OCA-eligible but not currently OCA-treated)

- Meet PBC claims diagnostic criteria (1 inpatient or 2 outpatient claims)
- Have at least 270 days of UDCA use before elevated ALP and/or TB inclusive of up to 4 instances of elevation (inadequate response) or <90 days UDCA use despite elevated ALP and/or bilirubin (intolerant)
- Have elevated ALP >ULN and/or TB >ULN

The Komodo Health database has not yet been linked to LabCorp laboratory database. It is anticipated that the number of patients in each group will approximately double with the availability of LabCorp data.

Global PBC registry: The Global PBC registry data are currently being refreshed. A previous analysis identified 344 patients who had initiated OCA. Among the >5000 patients not treated with OCA, it is anticipated that >2200 will meet criteria for UDCA failure and for inclusion in the control group (Corpechot 2008, Kumagi 2010).

#### **Diagnosis and Main Criteria for Inclusion:**

The treatment group will be patients with PBC with a history of inadequate response or intolerance to UDCA who initiated OCA in the study window. The control group will be PBC patients with a history of inadequate response or intolerance to UDCA who were eligible but not treated with OCA (or off-label fibrates) in the study window.

#### **Key Inclusion Criteria**

A patient who meets all of the following criteria for a given index date is eligible for inclusion:

- Definite or probable PBC diagnosis
  - o Global PBC registry (consistent with American Association for the Study of Liver Diseases [AASLD] and the European Association for the Study of the Liver [EASL] practice guidelines; Lindor 2009, EASL 2009): presence of ≥2 of the following 3 diagnostic factors:
    - History of elevated ALP levels for at least 6 months
    - Positive antimitochondrial antibody (AMA) titer
    - Liver biopsy finding consistent with PBC
  - o Komodo Health claims data: one of the following (Meyers 2010):
    - ≥1 inpatient claim with a PBC admission diagnosis at any position (ie, primary, secondary diagnosis, etc.)
    - ≥2 outpatient claims with a PBC diagnosis on separate days
- Inadequate response or intolerant to UDCA (see definitions below)
- Age  $\geq$ 18 years at the index date
- Continuous enrollment and evaluable data for at least 12 months before the index date (inclusive)

# **Key Exclusion Criteria:**

A patient who meets **any** of the following criteria for a given index date is not eligible for inclusion:

- History or presence of the following concomitant liver diseases before the index date (inclusive), including:
  - Acute or chronic hepatitis C virus infection
  - o Acute or chronic hepatitis B infection
  - Primary sclerosing cholangitis
  - Active alcoholic liver disease
  - Hepatocellular carcinoma
  - Hepatorenal syndrome
  - Hepatopulmonary syndrome
  - Portopulmonary syndrome
  - o Nonalcoholic steatohepatitis (NASH)
- History of non-skin malignancy or melanoma before the index date (inclusive)
- History of HIV before the index date (inclusive)
- Medical conditions that may cause non-hepatic increases in ALP such as:
  - o Paget's disease during the 12-month period before the index date (inclusive)
  - Fractures within 3 months before the index date (inclusive)

 Patients with laboratory values indicative of hepatic decompensation or significant hepatobiliary injury before the index date (inclusive)

- $\circ$  TB >3 mg/dL
- o ALP >10x ULN
- ALT and/or AST >10x ULN
- History of liver transplant before the index date (inclusive)
- Evidence of OCA, fenofibrate, or bezafibrate use before the index date (inclusive)
- History or presence of any of the following hepatic decompensating events before the index date (inclusive):
  - Variceal bleeding
  - Ascites
  - Hepatic hydrothorax
  - Spontaneous bacterial peritonitis
  - O Hepatic encephalopathy

#### **Definitions:**

- UDCA failure:
  - o Inadequate response requires both of the following:
    - At least 1 measure of ALP>ULN and/or TB>ULN
    - >270 days of UDCA treatment prior to ALP and/or TB elevation
  - Intolerant:
    - A maximum of 90 days of UDCA use with ALP>ULN and/or TB >ULN

#### **Group Assignments:**

- Treatment group (OCA-treated): ≥1 prescription or medical claim for OCA at or after UDCA failure date. The first date will be the one index date.
- Control Group (Non-OCA-treated but eligible for OCA): Each date corresponding to evidence of a patient meeting the definition of UDCA inadequate response or intolerance in which the patient meets the inclusion and exclusion criteria and does not initiate OCA will be an index date for the non-OCA-treated patient group. Patients may contribute indices to this group before they initiate OCA, but not after OCA index.

# Study medication, Dosage and Mode of Administration:

OCA tablet, 5 mg to 10 mg, once daily, oral administration

Patients may down titrate to <5 mg daily, but are censored if dose exceeds 10 mg per day.

Study drug is not provided nor administered by the Sponsor but is recorded by either administrative claim or registry CRF.

Duration of treatment will range from 1 to 67 months

# Reference Therapy, Dosage and Mode of Administration:

Not applicable

#### **Data Sources**

The data source for each analysis will include one of the following:

- 1. Komodo Health US administrative claims database linked to the following:
  - Laboratory measures (Quest Diagnostics and LabCorp)
  - National Death Index (US NDI)
  - National transplant registry (OPTN registry)

Or

Global PBC registry

#### **Criteria for Evaluation:**

#### Primary Outcome:

As-treated time to the first event of the composite endpoint of all-cause death, liver transplant, or hospitalization for hepatic decompensation, whichever occurs first.

#### **Exploratory Outcomes:**

As-treated time to the first occurrence of individual components of the composite endpoint:

- All-cause death
- Liver transplant
- Hepatic decompensation requiring hospitalization assessed through claims or registry CRF and defined as first occurrence of:
  - Variceal bleed
  - Ascites (including hepatic hydrothorax and spontaneous bacterial peritonitis)
  - o Hepatic encephalopathy

#### Exposure Variable:

The exposure variable is the use of OCA initiated at the index date.

#### Covariates:

The following covariates/control variables will be assessed **in the pre-index period**, utilizing the value closest to the index date:

- Age at index date
- Sex
- Most recent liver biochemistry levels (TB, ALP, ALT, AST)
- Most recent platelet counts
- Time (in months) since UDCA failure
- Clinical evidence of portal hypertension (platelets <150,000 and/or non-bleeding varices)
- Cirrhosis
- Most recent Charlson Comorbidity Index Score
- Insurance type at index date (Komodo Health only)

#### **Statistical Methods:**

#### **Analysis Populations**

The statistical analysis of the HEROES PBC studies will follow a nested randomized trial emulation approach (Hernán 2008, Danaei 2013) using a treatment decision design to identify index events (Brookhart 2015). Due to the lack of randomization, non-randomized observational studies will instead be conducted, with the goal of mimicking the hypothetical randomized trial as closely as possible. All patients will be evaluated over time from the start of the study period to identify evidence of inadequate treatment response to UDCA. Each date of inadequate response identified in the data will be considered a treatment decision point, and that date will be considered an index date, with a corresponding record created in the analytic data for that patient index. Each patient can contribute multiple index dates and thus patient indices, corresponding to each date they have a treatment decision point, and therefore each patient may contribute person-time to multiple patient index records.

It is likely that OCA-treated and non–OCA-treated patient indices will differ on confounding variables, ie, variables that influence both treatment and outcome. To address differences in the covariate distribution between treatment groups, the Sponsor will first conduct descriptive analyses on all baseline variables (demographics, clinical characteristics, and treatment history) for the OCA-treated and non–OCA-treated groups at index. Standardized mortality/morbidity ratio (SMR) weights then will be used to create a pseudo-population of non–OCA-treated indices with the same covariate distribution as the OCA-treated patients at the time of OCA initiation (Sato 2003), and unweighted and weighted standardized mean differences will be computed.

#### **Primary Analysis:**

The objective of the primary analysis is to estimate the as-treated effect of OCA treatment versus non–OCA-based treatment on the composite endpoint of all-cause death, liver transplant, or decompensation requiring hospitalization. The primary analysis outcome will be assessed with the hazard ratio comparing the hazard of the first event of the composite endpoint among the OCA-treated patients and standardized morbidity ratio-weighted

non—OCA-treated PBC patient indices. The hazard ratio will be estimated using a Cox proportional hazards model. The nonparametric bootstrap will be used to estimate the standard error of the estimate, which will then be used to generate 95% CI for the hazard ratio and to perform a test of the hypothesis that the hazard ratio is equal to the null value of 1.

## **Exploratory Analysis:**

The exploratory objectives are to estimate the effect of OCA treatment versus non-OCA treatment on each component of the composite endpoint (all-cause death, liver transplant, or hepatic decompensation). The exploratory analysis outcomes will be assessed with the subdistribution hazard ratio comparing the hazard of the first event of each element of the composite endpoint, separately, among the OCA-treated patients and standardized morbidity ratio-weighted non-OCA-treated PBC patient indices. For the endpoint of liver transplant, death will be treated as a competing event. For the endpoint of hepatic decompensation, death and liver transplant will be treated as competing events. The subdistribution hazard ratio will be estimated using a Fine-Gray proportional subdistribution hazards model. The nonparametric bootstrap will be used to estimate the standard error of the estimates, which will then be used to calculate 95% CI for the hazard ratio and perform a test of the hypothesis that the hazard ratio is equal to the null value of 1.

# Sample Size Justification:

Using the expected sample size in the 2 populations, the Sponsor computed power to detect treatment effects (relative hazards) of varying sizes, estimated using Cox proportional hazards regression. Computations are based on the formulae of Schoenfeld 1983. To account for confounding control due to the application of IP weights, the Sponsor inflated the variance from the Schoenfeld formula using factors derived by Shook-Sa 2020. It was conservatively assumed just one control observation per patient. In the Komodo Health data, a preliminary investigation found that approximately 395 patients who meet entry criteria initiate OCA and that 5916 patients will contribute at least one record to the control group (UDCA nonresponders). In the Global PBC registry, the Sponsor expects to have 344 patients meeting entry criteria who initiate OCA, and 2200 who contribute at least one observation to the control group. Power in both cohorts was computed for relative hazards ranging from 0.5 to 0.9 with an alpha level of 0.05. The Sponsor considered baseline event rates during follow-up from 5% to 15% and variance inflation corresponding to mild confounding (VIF=1.05), moderate confounding (VIF=1.5), and strong confounding (VIF=2.0). In each study, power was plotted under these assumptions against a reference line of 80% power under moderate confounding (VIF=1.5).

Under mild confounding, both studies will be well-powered to detect an HR of 0.5. For moderate confounding, the Komodo Health study will be adequately powered to detect HR of 0.5 for event rates >6%. The Global PBC registry will be adequately powered to detect event rates >8%. Under strong confounding, the Komodo Health study will be adequately powered to detect HR of 0.5 for event rates >9%. The Global PBC registry will be adequately powered to detect event rates >11%. Power decreases for more moderate HRs. None of the studies under even the most favorable assumptions will be able to detect HRs of 0.9. The Sponsor notes that the assumptions made here are conservative; in particular, it is expected that many more than one control observation and that the addition of lab data from LabCorp to will substantially increase the size of both treatment groups in the Komodo Health study.

# **Subgroup Analyses:**

The entire analysis will be repeated separately by patient race (Komodo Health only), age (categorical), sex, region, presence/absence of cirrhosis, and pre-/post-COVID. Because race is not completely captured in either database, these analyses will only include those with non-missing values for race.

#### **Sensitivity Analyses:**

- An analysis will be conducted in the Komodo database to assess the performance of a claims-based PBC definition with AMA test results as the gold standard.
- Quantitative bias analysis to quantify the sensitivity of the estimate to violations of the assumption of no unmeasured confounding.

# 2. TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES

# TABLE OF CONTENTS

| 1. | SYNOPSIS | 5 |
|--------|--------------------------------------------------------|----|
| 2. | TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES | 11 |
| 3. | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 14 |
| 4. | INTRODUCTION | 16 |
| 4.1. | Overview of Disease State and OCA | 16 |
| 4.2. | Mechanism of Action of OCA | 16 |
| 4.3. | Nonclinical Experience with OCA | 17 |
| 4.4. | Clinical Experience with Obeticholic Acid | 17 |
| 4.5. | Rationale for Study Design and Dose for OCA | 19 |
| 4.5.1. | Rationale for Study Design | 19 |
| 4.5.2. | Rationale for Dose | 19 |
| 4.5.3. | Rationale for Control Group | 19 |
| 4.6. | Summary of Safety with OCA | 19 |
| 4.6.1. | Clinical Trial Exposure and Safety Experience | 19 |
| 4.6.2. | Known and Potential Risks of OCA | 20 |
| 5. | STUDY OBJECTIVES AND PURPOSE | 22 |
| 5.1. | Primary Objective | 22 |
| 5.2. | Exploratory Objectives | 22 |
| 6. | INVESTIGATIONAL PLAN | 22 |
| 6.1. | Overall Design | 22 |
| 6.1.1. | Design Diagram | 23 |
| 6.2. | Number of Patients | 23 |
| 7. | SELECTION OF PATIENTS | 24 |
| 7.1. | Study Population. | 24 |
| 7.1.1. | Definition of UDCA Failure | 24 |
| 7.2. | Inclusion Criteria | 25 |
| 7.3. | Exclusion Criteria | 25 |
| 7.4. | Group Assignments | 26 |
| 7.5. | Study Product, Dosage and Mode of Administration | 27 |

| 7.6. | Study Period | 27 |
|---------|-------------------------------------------|----|
| 8. | ASSESSMENT OF EFFICACY | 27 |
| 8.1. | Primary Outcomes/Endpoints | 27 |
| 8.2. | Exploratory Outcomes | 29 |
| 8.3. | Exposure Variable | 29 |
| 9. | ASSESSMENT OF SAFETY | 29 |
| 10. | STATISTICAL METHODS | 29 |
| 10.1. | Analysis Populations and Blinding | 29 |
| 10.1.1. | Analysis Populations | 29 |
| 10.1.2. | Blinding | 32 |
| 10.2. | Estimation of Effect Size | 32 |
| 10.3. | Hypotheses | 33 |
| 10.3.1. | Primary Hypothesis | 33 |
| 10.4. | Determination of Sample Size | 33 |
| 10.5. | Primary Efficacy Analysis | 34 |
| 10.6. | Exploratory Analyses | 35 |
| 10.7. | Handling of Dropouts or Missing Data | 35 |
| 10.8. | Subgroup Analyses | 35 |
| 10.9. | Sensitivity Analyses | 35 |
| 10.10. | Assessment of Claims-based PBC Definition | 36 |
| 10.11. | Clean Room Committee | 36 |
| 11. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 37 |
| 12. | QUALITY CONTROL AND QUALITY ASSURANCE | 38 |
| 12.1. | Data Collection and Transfer | 38 |
| 12.1.1. | Komodo Health | 38 |
| 12.1.2. | Global PBC Registry | 38 |
| 12.1.3. | National Death Index | 39 |
| 12.1.4. | Quest Diagnostics | 39 |
| 12.1.5. | LabCorp | 39 |
| 12.1.6. | OPTN Transplant Registry | 39 |
| 12.2. | Data De-identification | 40 |
| 12.2.1. | Global PBC Registry | 40 |

| 12.2.2. | Komodo Health | 40 |
|---|---|---|
| 12.3. | Data Linkages | 41 |
| 12.4. | Data Harmonization | 42 |
| 12.4.1. | Komodo Health and National Death Index | 42 |
| 12.4.2. | Komodo Health and OPTN Liver Transplant | 42 |
| 12.4.3. | Komodo Health Hospitalization for Hepatic Decompensation | 42 |
| 12.4.4. | Quest Diagnostics and LabCorp | 43 |
| 12.4.5. | Cirrhosis | 44 |
| 12.5. | Characterization of Missing Data | 46 |
| 12.6. | Data Management and Analysis SOPs | 46 |
| 12.7. | Audits and Inspections | 46 |
| 12.8. | Quality Control and Quality Assurance | 46 |
| 12.9. | Data Retention and Archiving Study Documents | 46 |
| 13. | PROTECTION OF HUMAN SUBJECTS | 47 |
| 14. | ADVERSE EVENT REPORTING | 47 |
| 15. | PUBLICATION POLICY | 47 |
| 16. | LIST OF REFERENCES | 49 |
| APPENDI | X A. LIST OF INCLUSION, EXCLUSION AND COVARIATE CODES | 51 |
| APPENDI | X B. TABLE SHELLS | 70 |
| | LIST OF TABLES | |
| Table 1: | Composite Endpoints for OCA PBC Studies | 28 |
| Table 2: | Comparison of Imaging-based (Global PBC) and Claims-based (HealthCore, Optum) Prevalence of Cirrhosis in PBC Patients. | |
| | LIST OF FIGURES | |
| Figure 1: | Design Schematic Studies 747-404/405 | 23 |
| Figure 2: | Power estimates by Hazard Ratio by Level of Confounding for Komodo Health (A) and Global PBC Registry (B). | 34 |
| Figure 3: | Incidence Rates for Major Hepatic Events Stratified by Cirrhosis, Portal Hypertension and Hepatic Decompensation in the Optum (A) and HealthCore (B) Databases | 45 |

# 3. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

The following abbreviations and specialist terms are used in this protocol.

| Abbreviation or Specialist Term | Explanation |
|---|---|
| AASLD | American Association for the Study of Liver Diseases |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| AMA | antimitochondrial antibody |
| AST | aspartate aminotransferase |
| CDCA | chenodeoxycholic acid |
| CRC | Clean Room Committee |
| CRO | Clinical Research Organization |
| CVD | cardiovascular disease |
| DB | double-blind |
| DMC | data monitoring committee |
| EASL | European Association for the Study of the Liver |
| eCRF | electronic case report form |
| EU | European Union |
| FDA | Food and Drug Administration |
| FXR | farnesoid X receptor |
| ICD | International Classification of Diseases |
| ICMJE | International Committee of Medical Journal Editors |
| IEC | Independent Ethics Committee |
| IRB | Institutional Review Board |
| HIPAA | Health Insurance Portability and Accountability Act |
| INR | international normalized ratio |
| ITT | intent-to-treat |
| LLN | lower limit of normal |
| LTSE | long-term safety extension |
| MELD | Model for End-Stage Liver Disease |
| NASH | nonalcoholic steatohepatitis |
| NDI | National Death Index |
| OCA | obeticholic acid |
| OPTN | Organ Transplant Network |

| Abbreviation or Specialist Term | Explanation |
|---------------------------------|----------------------------------|
| PBC | primary biliary cholangitis |
| PD | pharmacodynamic(s) |
| PK | pharmacokinetic(s) |
| PPV | positive predictive value |
| QD | once per day |
| RWE | real-world evidence |
| SDTM | Study Data Tabulation Model |
| SMD | standardized mean differences |
| SOP | standard operating procedure |
| ТВ | total bilirubin |
| TEAE | treatment-emergent adverse event |
| UDCA | ursodeoxycholic acid |
| ULN | upper limit of normal |
| US | United States |

# 4. INTRODUCTION

# 4.1. Overview of Disease State and OCA

Primary biliary cholangitis, (PBC) is a serious, life-threatening, cholestatic liver disease of unknown etiology that, without treatment, frequently progresses to hepatic fibrosis and eventual cirrhosis or hepatic decompensation and necessitates liver transplantation or results in death. PBC is a rare disease with a reported prevalence in the United States (US) of 40/100,000 (Kim 2000). PBC disproportionately affects women (with a female to male ratio of approximately 10:1) and is typically diagnosed in patients aged 40 to 60 years.

The only approved drug therapy for PBC has been the bile acid ursodeoxycholic acid (UDCA), a physiological constituent of human bile (Lindor 2009). While UDCA therapy had a marked effect on the treatment of PBC, up to 40% of patients showed a suboptimal response or no response to UDCA (Corpechot 2008, Kumagi 2010). Such patients were at significantly increased risk of a poor clinical outcome due to PBC disease progression. Obeticholic acid (OCA) is a farnesoid X receptor (FXR) agonist and a modified bile acid that is derived from the primary bile acid chenodeoxycholic acid (CDCA), the natural human FXR ligand. OCA (Ocaliva®) has received marketing authorization in the US, the European Union (EU), and several other countries for the treatment of PBC in combination with UDCA in adults with an inadequate response to UDCA or as monotherapy in adults unable to tolerate UDCA. In the US, Ocaliva is contraindicated in patients with decompensated cirrhosis (eg, Child-Pugh Class B or C), a prior decompensation event, complete biliary obstruction, or compensated cirrhosis with evidence of portal hypertension. Approval in the US and the EU was based on a surrogate endpoint (reduction in ALP), and as part of regulatory commitments in these regions, the following postmarketing studies were initiated: Study 747-302, a Phase 3b/4 study designed to prospectively obtain evidence to confirm clinical benefit in PBC subjects, and Study 747-401, a Phase 4 study designed to evaluate the pharmacokinetics (PK) and safety of OCA in PBC subjects with hepatic impairment. Both 747-302 and 747-401 terminated early, due to the challenges of recruitment and long-term retention of patients with a rare disease subsequent to Ocaliva regulatory approval. Changes to endpoints and statistical analysis plans to accommodate low recruitment, low events rates, and early termination may necessitate the need for clinical trial data to be supplemented with real-world evidence, with the goal of providing regulators with a more complete evidence package characterizing the efficacy and safety of OCA in patients with PBC.

# 4.2. Mechanism of Action of OCA

OCA is a  $6\alpha$ -ethyl derivative of the naturally occurring primary human bile acid CDCA, which is the endogenous ligand for FXR. FXR is a ligand-dependent transcription factor that is part of the nuclear receptor superfamily. FXR regulates a wide variety of target genes involved in the control of bile acid, lipid, and glucose homeostasis and in the regulation of immune responses. OCA's potent FXR agonist effects are believed to account for the predominant efficacy of the investigational product. Some of the pharmacological properties of OCA and other FXR agonists that have been elucidated in animal models of chronic liver disease relevant to the treatment of PBC include the following:

• Improvement in hepatic choleresis with reduced inflammation and necrosis

• Prevention and reversal of hepatic fibrosis

The key mechanisms of action of OCA, including its choleretic, anti-inflammatory, and anti-fibrotic properties, underlie its hepatoprotective effects and result in attenuation of injury and improved liver function in a cholestatic liver disease, such as PBC.

# 4.3. Nonclinical Experience with OCA

Intercept Pharmaceuticals, Inc. (the Sponsor) has completed a standard battery of nonclinical safety pharmacology and toxicology studies. No major nonclinical safety effects have been seen other than pharmacologic hepatic effects observed at high doses. These pharmacologic hepatic effects are consistent with the detergent effects of a bile acid at exceedingly high hepatocellular exposure.

# 4.4. Clinical Experience with Obeticholic Acid

As of 03 May 2021, approximately 4438 subjects have received ≥1 dose of OCA. This estimation includes subjects from blinded ongoing studies. Of these subjects, 978 were healthy volunteers, 610 subjects had PBC, 72 subjects had primary sclerosing cholangitis, 7 subjects had biliary atresia, 41 subjects had diabetes mellitus with non-alcoholic fatty liver disease, 2697 subjects had nonalcoholic steatohepatitis (NASH), and 33 subjects had portal hypertension due to alcoholic cirrhosis.

As of 03 May 2021, the clinical pharmacology of OCA had been evaluated in 19 completed Phase 1 studies. Overall, the PK of OCA shows the profile expected of a natural bile acid. There is rapid absorption of unconjugated OCA (parent), followed by extensive conjugation to glycine and taurine to form glyco-OCA and tauro-OCA, respectively. Glyco-OCA and tauro-OCA occur at significantly higher concentrations than the parent drug does. There are numerous peak and trough plasma concentrations observed, consistent with the expected extensive enterohepatic circulation of a bile acid. Plasma concentrations dramatically increase shortly after food intake, consistent with the gall bladder emptying into the duodenum. The glyco-OCA and tauro-OCA conjugates of OCA are known to be pharmacologically active, and due to enterohepatic recycling of OCA and its conjugates, their plasma PK profiles are most relevant.

Data that supported approval of Ocaliva included 3 randomized, double-blind, placebo-controlled, multi-center, international studies in subjects with PBC:

- Study 747-201 was a Phase 2, 3-month, international, double-blind, placebo-controlled, parallel-group study in subjects with a proven or likely diagnosis of PBC whose disease was sub-optimally controlled. In this study, OCA doses of 10 mg and 50 mg were evaluated as monotherapies.
- Study 747-202 was a Phase 2, 3-month, international, double-blind, placebo-controlled, parallel-group study in subjects with a proven or likely diagnosis of PBC who were sub-optimally controlled. OCA doses of 10 mg, 25 mg, and 50 mg were evaluated as add-on therapy to UDCA, the current standard of care for PBC.

• Study 747-301(POISE) was the pivotal Phase 3, 12-month, international, double-blind, placebo-controlled study in subjects with a proven or likely diagnosis of PBC whose disease was sub-optimally controlled. In this study, OCA doses evaluated were 10 mg or a titration approach (ie, 5 mg for the initial 6 months, with up-titration to 10 mg for the last 6 months if the subject did not meet the primary composite endpoint and had no tolerability issues).

In the double-blind, Phase 2 Studies 747-201 and 747-202, treatment with OCA for 3 months in subjects with PBC resulted in statistically and clinically significant reductions in ALP, a known surrogate for risk of long-term clinical outcomes in PBC, as well as markers of hepatic damage and inflammation. Consistent efficacy results were observed irrespective of whether OCA was administered as monotherapy or as an add-on to UDCA. Within each study, OCA doses above 10 mg did not show substantially better efficacy compared with OCA 10 mg, but the incidence and severity of pruritus were increased, suggesting that 10 mg was the maximally efficacious dose and that evaluation of lower doses in the Phase 3 program was warranted.

The Phase 3 study met its primary endpoint. Both OCA treatment groups (OCA titration and OCA 10 mg) were superior to placebo in achieving the primary endpoint at all timepoints across the 12-month treatment period (p<0.0001 versus placebo).

Each of these 3 studies included open-label, uncontrolled, long-term safety extension (LTSE) phases to evaluate the long-term effects of OCA treatment. As of 03 May 2021, the LTSEs of Studies 747-201, 747-202, and 747-301 are completed.

Study 747-301 LTSE: A total of 217 subjects were enrolled into the double-blind phase of the study; of the 198 subjects who completed the double-blind phase, 193 subjects (98%) enrolled into the LTSE phase. Overall, there was good retention in the study: 146 (76%) subjects completed the protocol as specified after administrative termination/closure of the study, and 47 (24%) subjects discontinued the LTSE prematurely. The majority of subjects discontinued because of study closure by the Sponsor. The efficacy associated with continued treatment with OCA up to 6 years was durable and consistent with the effects observed in the double-blind phase.

An additional 8-week, open-label study was also supportive of Ocaliva approval; however, efficacy data from this study were not integrated with Studies 747-201, 747-202, and 747-301 because of differences in study design and endpoints:

• Study 747-205 assessed the safety, tolerability, and pharmacodynamic (PD) effects of OCA on high-density lipoprotein cholesterol metabolism in subjects with PBC on a stable dose of UDCA. The LTSE phase is considered complete the clinical study report approved 07 Jan 2021.

Postmarketing studies in subjects with PBC include the following:

• Study 747-302 (COBALT; postmarketing requirement) is a double-blind, randomized, placebo-controlled, multicenter study designed to prospectively obtain evidence to confirm clinical benefit and further evaluate the benefit-risk profile of OCA treatment in subjects with PBC. Last Patient Last Visit occurred on 23 Dec 2021.

 Study 747-401 (postmarketing requirement) is a double-blind, randomized, placebo-controlled study evaluating the PK and safety of OCA in subjects with PBC and moderate to severe hepatic impairment. This study was closed as of 09 Jul 2021.

# 4.5. Rationale for Study Design and Dose for OCA

# 4.5.1. Rationale for Study Design

Studies 747-404 and 747-405 are replicate, observational, retrospective cohort studies. In rare diseases, real-world retrospective observational studies utilizing claims and registry data have been recognized by the US Food and Drug Administration (FDA) as viable for various regulatory use-cases, including constructing of external control arms for clinical trials (US Food and Drug Administration 2018, US Food and Drug Administration 2021).

The analytic approach, a nested randomized trial emulation using a treatment decision design to identify index events (Hernán 2008, Danaei 2013, Brookhart 2015), was selected to best mimic a clinical trial and has been shown to replicate trial results in epidemiologic data when other real-world approaches have not (Hernán 2008). This design emulates a sequence of hypothetical randomized trials, and, though non-randomized and non-blinded, mimics trial eligibility criteria, definition of start of follow-up, and treatment arms (initiators vs. non-initiators). Standardized morbidity ratio-weighting is used to adjust for imbalances in patient characteristics at index. The approach will produce an average hazard (rate) ratio (HR) and 95% confidence interval, comparing OCA initiators to non-initiators, thus yielding the standard output of a clinical study that is amenable to statistical hypothesis testing (ie, null hypothesis: HR=1). An as-treated approach was deemed superior to an intent-to-treat (ITT) approach, as the ITT approach in epidemiological data often causes severe treatment misclassification, particularly in chronic disease (Hernán 2008).

#### 4.5.2. Rationale for Dose

The Ocaliva prescribing information states that the approved dosing is 5 mg once daily (QD) with allowable up-titration to a maximal dose of 10 mg QD. Patients prescribed OCA will be censored if they exceed the maximal allowable daily dose. Down-titration (less than daily dosing) can be utilized in response to adverse events such as pruritus, and as such, patients dosed <5 mg QD will continue to be counted in the OCA-treated arm.

# 4.5.3. Rationale for Control Group

Using standardized eligibility criteria across treated and untreated patients and utilizing a standardized morbidity ratio—weighted-OCA eligible but non—OCA-treated comparator group will provide the best scientific comparative evidence of efficacy.

# 4.6. Summary of Safety with OCA

# 4.6.1. Clinical Trial Exposure and Safety Experience

As of 03 May 2021, approximately 6183 subjects have been enrolled in the development program for OCA. Approximately 4438subjects received ≥1 dose of OCA in clinical studies sponsored by Intercept and Sumitomo Dainippon Pharma Co., Ltd. (Intercept's former

development partner in China, Korea, and Japan). Of these, a total of 610 PBC subjects had received ≥1 dose of OCA in completed (Studies 747-201 Double-Blind [DB], 747-201 LTSE, 747-202 DB, 747-202 LTSE, 747-205 Primary Treatment Phase, 747-301 DB, and 747-301 LTSE), ongoing unblinded (Study 747-205 LTSE), or blinded (Studies 747-302 and 747-401) studies.

In the completed studies, the majority of subjects had at least 5 years of exposure to OCA, and a small subset were exposed for more than 7 years. A total of 421 (97%) of these subjects who received OCA experienced treatment-emergent adverse events (TEAEs) during the study, and 379 (88%) subjects experienced investigational product—related TEAEs. Although the rate of TEAEs was higher in OCA-treated subjects compared with placebo-treated subjects, the differences noted in these incidence rates may be at least partially due to cumulative exposure differences between OCA and placebo. The most frequently reported TEAEs by System Organ Class in subjects receiving OCA were those classified as skin and subcutaneous tissue disorders (84%), gastrointestinal disorders (62%), and infections and infestations (56%). The most frequently reported (≥20% of subjects) individual TEAEs were pruritus (80%) and fatigue (26%).

While studies were ongoing, the data monitoring committee (DMC) convened at least every 6 months to review safety data for ongoing, double-blind, placebo-controlled postmarketing requirement studies 747-302 and 747-401. On 25 Mar 2020, the DMC recommended that both studies continue without modifications, consistent with prior periodic reviews. On 28 Sep 2020, the DMC reviewed a planned interim efficacy analysis for Study 747-302. The DMC noted that based on their review, they did not have additional analyses to suggest to better understand the observed hazard rate. They also noted that it did not seem feasible to continue the study as designed. On 18 Dec 2020, the DMC reviewed a planned in-depth analysis of unblinded safety data from Studies 747-302 and 747-401. Enrollment and retention were particularly poor in Study 747-302 in subjects with decompensated cirrhosis at baseline. Poor retention was also observed in Study 747-401, which is exclusively focused on subjects with CP-B and CP-C cirrhosis at baseline. The DMC noted a high likelihood of futility and difficulty in differentiating the etiology of hepatic safety events (OCA-related or progression of underlying disease). No safety concerns were raised by the DMC for either study. The DMC recommended stopping further enrollment in Studies 747-302 and 747-401 and discussing the unblinding of both studies with regulators. On 17 Feb 2021, the DMC recommended that both studies continue with modification. Due to the high likelihood of futility, the DMC recommended no further enrollment in the studies. On 09 Jun 2021, no additional modifications to the study were recommended. The DMC's previous recommendations remained unchanged (ie, continue discussion with regulatory authorities regarding unblinding). Following the United States Prescribing Information update on 26 May 2021, Study 747-401 was closed as of 09 Jul 2021. On 03 Nov 2021, after careful consideration of feedback from the DMC and the FDA, Intercept terminated Study 747-302 with Last Patient Last Visit completed on 23 Dec 2021.

# 4.6.2. Known and Potential Risks of OCA

The risk profile of OCA use in PBC has been evaluated in clinical trials and observational studies, as well as from postmarketing experience (estimated cumulative patient exposure from marketing experience is 20,554 patient-years). The key risk for OCA is pruritus. Potential risks

include liver injury and atherosclerotic cardiovascular events secondary to changes in lipids. The following focuses on these risks in the context of PBC, the subject of these current studies. Additional information is available in the Investigator's Brochure.

Pruritus: In subjects with PBC, the most commonly reported TEAE across all treatment groups was pruritus, which is a frequent symptom experienced by subjects with cholestatic liver disease. The incidence of pruritus was higher in the OCA-treated subjects as compared with placebo-treated subjects. In a small proportion of patients, pruritus can be severe and significantly interfere with sleep and patient functioning. Patients with a history of pruritus as part of the underlying disease have a higher probability of pruritus with OCA treatment. Otherwise, the occurrence and severity of pruritus in an individual patient treated with OCA cannot be reliably predicted or prevented, in part because pruritus is a frequent clinical feature of the underlying disease. Pruritus has also been seen in patients participating in clinical trials of investigational use of OCA, including NASH, where pruritus is not a common symptom of the disease state. Pruritus is generally clinically manageable. Reducing OCA dose or transient dose or transient treatment interruption helps alleviate, and in some cases, even resolves it.

<u>Liver Injury</u>: Liver injury is an important potential risk for OCA. Risk factors for drug-induced adverse hepatic effects are in general poorly understood in patients with chronic liver disease. Pre-existing liver disease may not increase the risk of developing drug-induced liver injury (Chalasani 2014). In the US, OCA is contraindicated in adult patients with PBC with decompensated cirrhosis or a prior decompensation event and with compensated cirrhosis with clinical evidence of portal hypertension. OCA is also contraindicated in adult patients with PBC with complete biliary obstruction.

In two 3-month, placebo-controlled studies in subjects with PBC, a dose-response was observed for the occurrence of liver-related adverse reactions including jaundice, worsening ascites, and PBC flare with dosages of OCA 10 mg to 50 mg once daily (up to 5-times the highest recommended dosage in PBC). In a pooled analysis of 3 placebo-controlled studies in subjects with PBC, the exposure-adjusted incidence rates for all serious and otherwise clinically significant liver-related adverse reactions and isolated elevations in liver biochemical tests, per 100 patient years of exposure were: 5.2 in the OCA 10 mg group, 19.8 in the OCA 25 mg group, and 54.5 in the OCA 50 mg group compared to 2.4 in the placebo group.

Atherosclerotic Cardiovascular Events Secondary to Changes in Lipids: This risk has been recognized as an important potential risk since OCA is associated with lipid profile changes, regardless of background disease state. Patients with PBC generally exhibit hyperlipidemia characterized by a significant elevation in total cholesterol. A reduction in mean high-density lipoprotein and an increase in low-density lipoprotein with OCA treatment have been observed in patients with PBC. It is unknown whether these changes in lipids are associated with or are causally related to an increased risk of atherosclerotic cardiovascular disease (CVD) and associated morbidity and mortality in PBC patients, when compared with the general population. The lipid abnormalities may be managed in PBC patients receiving OCA, by monitoring and managing lipid levels and other CVD risk factors.

# 5. STUDY OBJECTIVES AND PURPOSE

The overall objective of these studies is to evaluate the effectiveness of OCA on hepatic outcomes in patients with PBC who failed UDCA treatment in 2 real-world data sources: Global PBC registry and Komodo Health claims database.

# 5.1. Primary Objective

To evaluate the effect of OCA treatment on time to the first occurrence of the composite endpoint of all-cause death, liver transplant, or hospitalization for hepatic decompensation in PBC patients in 2 data sources: Global PBC registry and Komodo Health US claims database.

# 5.2. Exploratory Objectives

To evaluate the effect of OCA treatment on time to the first occurrence of individual components of the composite endpoint (outlined below):

- All-cause death
- Liver transplant
- Hospitalization for hepatic decompensation based on first occurrence of:
  - Variceal bleed
  - Ascites (including hepatic hydrothorax and spontaneous bacterial peritonitis)
  - Hepatic encephalopathy

# 6. INVESTIGATIONAL PLAN

# **6.1.** Overall Design

These are replicate, observational, retrospective cohort studies of patients with PBC who failed UDCA treatment using 2 real-world data sources: the Global PBC registry (Study 747-404) and the Komodo Health US claims database (Study 747-405). All analyses will be conducted separately by data source (ie, not pooled). The Komodo Health database will be linked for outcome verification and additional data collection through Datavant tokenization to Quest Diagnostics, LabCorp, the NDI, and the Organ Transplant Network (OPTN) registry.

All patients who meet diagnostic criteria for PBC in each database between 01 Jun 2015 and 31 Dec 2021 and who meet the eligibility criteria (Section 7.2 and Section 7.3) will be considered for these studies. See Figure 1 for the design schematic. The OCA treatment evaluation period will be from 01 Jun 2016 (based on first country approval by FDA on 27 May 2016). The Komodo Health database is US-specific, while the Global PBC registry includes multiple countries with a range of approval dates. The Sponsor has applied the date of first approval of a participating country, and thus 01 Jun 2016 will be used for both studies. The first date of prescription of OCA after failing UDCA treatment will be defined as the index date for OCA-treated PBC patients. The date of evidence of inadequate UDCA response or UDCA intolerance, as defined in Section 7.1, will be used as an index date for the non–OCA-treated comparator group. Each time a patient meets the UDCA inadequate response/intolerance

definition or the definition of OCA initiation, as well as all other inclusion criteria, they will contribute an index to the study. Therefore, patients may contribute multiple control indices, and may contribute control indices before OCA initiation, but can contribute only one OCA initiation index. The non–OCA-treated patient indices will be weighted to have the same baseline covariate distribution as the OCA-treated patients at the time of OCA initiation, thus allowing for the estimation of the effect of treatment in the treated. Patients must have 12 months of data preceding the index date (ie, the pre-index period) to establish the medical history and OCA eligibility and for the standardized morbidity ratio-weighting. Follow-up of patients will be until the first occurrence of the composite endpoint. Patients will be censored at drop out/disenrollment from the database, discontinuation of OCA (+90 days), initiation of fenofibrate or bezafibrate, initiation of OCA (for the non–OCA-treated patient indices), unapproved OCA dose (>10 mg QD) for those treated with OCA, or the end of the study period (31 Dec 2021); whichever comes first.

# 6.1.1. Design Diagram

Figure 1: Design Schematic Studies 747-404/405



# **6.2.** Number of Patients

The Komodo Health database contains administrative claims from >350 US payers, tokenized to allow for patient tracking across payers. Komodo Health claims will be linked through Datavant tokenization to Quest Diagnostics and LabCorp laboratory data, the US National Death Index (NDI), and the Organ Transplant Network (OPTN) transplant registry for additional information and outcome verification. The database contains >100,000 patients with a PBC diagnostic code. The Global PBC registry includes >5,000 patients with PBC recruited from 17 liver centers across 8 countries in Europe and North America. It utilizes the CASTOR trial platform for

electronic case report form (eCRF) collection of medical history, clinical events, and laboratory and treatment data.

<u>Komodo Health</u>: In the current Komodo Health database, there are 395 patients who meet criteria for the OCA treatment group:

- Meet PBC claims diagnostic criteria (1 inpatient or 2 outpatient claims)
- Initiate OCA treatment
- Have evidence of UDCA failure

There are 5916 who meet criteria for the control group (OCA-eligible but not currently OCA-treated)

- Meet PBC claims diagnostic criteria (1 inpatient or 2 outpatient claims)
- Have at least 270 days of UDCA use before elevated ALP and/or TB inclusive of up to 4 instances of elevation (inadequate response) or ≤90 days UDCA use before elevated ALP and/or TB (intolerant)
- Have evidence of ALP >ULN and/or TB >ULN

The Komodo Health data have not yet been linked to LabCorp laboratory data. It is anticipated that these numbers will approximately double with the availability of LabCorp data.

Global PBC Registry: The Global PBC registry data are currently being refreshed. A previous analysis identified that 344 patients who had initiated OCA. Among the >5000 patients not treated with OCA, it is anticipated that >2200 will meet criteria for UDCA failure and for inclusion in the control group (Corpechot 2008, Kumagi 2010).

# 7. SELECTION OF PATIENTS

# 7.1. Study Population

All patients who meet diagnostic criteria in each database between 01 Jun 2015 and 31 Dec 2021 and who meet the eligibility criteria will be considered for these studies.

All diagnosis, treatment, laboratory, and procedure codes used to identify patients and define study variables are listed in Appendix A.

The treatment group will be patients with PBC with a history of inadequate response or intolerance to UDCA who initiated OCA in the study window. The control group will be PBC patients with a history of inadequate response or intolerance to UDCA who were eligible but were not treated with OCA (or off-label fibrates) in the study window. The decision to treat a patient with OCA or UDCA is at the discretion of the treating physician and has been made independent from inclusion in each of the databases.

#### 7.1.1. Definition of UDCA Failure

UDCA failure includes both inadequate response to UDCA, and intolerance to UDCA. Inadequate UDCA response is defined as:

- At least 1 measure of ALP and/or TB >ULN; and
- $\geq$ 270 days of UDCA treatment prior to ALP and/or TB elevation

UDCA intolerance is defined as:

• A maximum of 90 days of UDCA use with ALP>ULN and/or TB >ULN.

The first date of prescription of OCA after inadequate UDCA response (ALP>upper limit of normal [ULN] and/or total bilirubin [TB]>ULN after >270 days of treatment) or UDCA intolerance (discontinued UDCA after <90 days despite ALP>ULN and/or TB>ULN) will be defined as the index date for OCA-treated PBC patients. The dates of evidence of inadequate UDCA response or UDCA intolerance during which OCA is not utilized will be used as index dates for the non–OCA-treated comparator group.

# 7.2. Inclusion Criteria

A patient who meets **all** of the following criteria for a given index date is eligible for inclusion:

- Definite or probable PBC diagnosis
  - Global PBC Registry (consistent with American Association for the Study of Liver Diseases [AASLD] and the European Association for the Study of the Liver [EASL] practice guidelines; Lindor 2009, EASL 2009): presence of ≥2 of the following 3 diagnostic factors:
    - History of elevated ALP levels for at least 6 months
    - Positive antimitochondrial antibody (AMA) titer
    - Liver biopsy finding consistent with PBC
  - Komodo Health claims data: one of the following (Meyers 2010):
    - ≥1 inpatient claim with a PBC admission diagnosis at any position (ie, primary, secondary diagnosis, etc.)
    - ≥2 outpatient claims with a PBC diagnosis on separate days
- Inadequate response or intolerance to UDCA (see definitions in Section 7.1)
- Age  $\geq$ 18 years at the index date
- Continuous enrollment and evaluable data for at least 12 months before the index date (inclusive)

# 7.3. Exclusion Criteria

A patient who meets **any** of the following criteria for a given index date is not eligible for inclusion:

- History or presence of other concomitant liver diseases before the index date (inclusive), including:
  - Acute or chronic hepatitis C virus infection
  - Acute or chronic hepatitis B infection

- Primary sclerosing cholangitis
- Active alcoholic liver disease
- Hepatocellular carcinoma
- Hepatorenal syndrome
- Hepatopulmonary syndrome
- Portopulmonary syndrome
- NASH
- History of non-skin malignancy or melanoma before the index date (inclusive)
- History of HIV before the index date (inclusive)
- Medical conditions that may cause non-hepatic increases in ALP:
  - Paget's disease during the 12-month period before the index date (inclusive)
  - Fractures within 3 months before the index date (inclusive)
- Patients with laboratory values indicative of hepatic decompensation or significant hepatobiliary injury before the index date (inclusive):
  - TB >3 mg/dL
  - ALP >10x ULN
  - ALT and/or AST >10x ULN
- History of liver transplant before the index date (inclusive)
- Evidence of OCA, fenofibrate, or bezafibrate use before the index date (inclusive)
- History or presence of any of the following hepatic decompensating events before the index date (inclusive):
  - Variceal bleeding
  - Ascites
  - Hepatic hydrothorax
  - Spontaneous bacterial peritonitis
  - Hepatic encephalopathy

# 7.4. Group Assignments

**Treatment group (OCA-treated)**: ≥1 prescription or medical claim for OCA at or after UDCA failure date. The first date will be the one index date.

Control Group (Non-OCA-treated but eligible for OCA): Each date corresponding to evidence of a patient meeting the definition of UDCA inadequate response or intolerance in which the patient meets the inclusion and exclusion criteria and does not initiate OCA will be an

index date for the non-OCA-treated patient group. Patients may contribute indices to this group before they initiate OCA, but not after OCA index.

A thorough description of methodology underlying group assignment can be found in Section 10.1.1.

# 7.5. Study Product, Dosage and Mode of Administration

The product being studied is obeticholic acid, in tablet form, dosed at 5 mg to 10 mg once daily oral administration. The study drug is not provided nor administered by the Sponsor but is recorded by either administrative claim or registry eCRF. The total duration of exposure will range from 1 to 67 months.

# 7.6. Study Period

The total study period is estimated to be a maximum of 6.6 years based on a pre-index period of 12 months prior to the index date and a maximum follow-up period of 5.6 years after the index date. The OCA treatment evaluation period will be from 01 Jun 2016 (based on FDA approval on 27 May 2016) to 31 Dec 2021. The first date of prescription of OCA after failing UDCA treatment will be defined as the index date for OCA-treated PBC patients. The date of evidence of inadequate UDCA response or UDCA intolerance, as defined below, will be used as the index date for the non–OCA-treated comparator group. Each time a patient meets the UDCA inadequate response/intolerance definition or the definition of OCA initiation, as well as all other inclusion/exclusion criteria, they will contribute an index to the study. Therefore, patients may contribute multiple indices and may appear in both groups, though they may contribute at most one index to the OCA-treated group.

# 8. ASSESSMENT OF EFFICACY

# 8.1. Primary Outcomes/Endpoints

The selection of a composite primary endpoint was informed by previous regulatory interactions regarding the 747-301 (POISE) and 747-302 (COBALT) studies (see Table 1). For COBALT, the primary composite endpoint included all-cause death, liver transplant, hospitalization for hepatic decompensation (bleeding varices and hepatic encephalopathy), uncontrolled ascites, and Model for End-Stage Liver Disease (MELD) Score ≥15. Of these endpoints, only MELD cannot be adequately assessed in the current databases. The MELD algorithm includes a measure of the international normalized ratio (INR). A review of the Komodo Health and the Global PBC registry databases revealed that, unlike hepatic laboratory measures such as ALP and TB, INR is not routinely collected in PBC patients. Therefore, the Sponsor did not include MELD ≥15 as part of the composite endpoint for these studies.

COBALT included the endpoint of uncontrolled ascites, defined as diuretic-resistant ascites requiring therapeutic paracentesis at a frequency of at least twice in a month. In a study of the POISE LTSE with external controls (Perez 2021), the Sponsor modified this endpoint to be consistent with other decompensating events, ie, hospitalization for ascites. As the FDA Guidance on Real-world Data (US Food and Drug Administration 2021) states, "...outpatient data sources that do not include hospitalization data would generally not be appropriate for studying outcomes likely to result in hospitalization." To increase consistency in the measures of

hepatic decompensating events, the Sponsor has included ascites (including hepatic hydrothorax and spontaneous bacterial peritonitis), along with variceal bleeding and hepatic encephalopathy, as part of the "hospitalization for hepatic decompensation" endpoint.

**Table 1:** Composite Endpoints for OCA PBC Studies

| | COBALT<br>(747-302) | POISE (747-301) LTSE with External Controls | HEROES PBC<br>(747-404/405) |
|---|---|---|---|
| All-cause death | X | X | X |
| Liver transplant | X | X | X |
| Hospitalization for hepatic decompensation Variceal bleed Hepatic encephalopathy | X | Х | Х |
| Uncontrolled ascites | X | X <sup>a</sup> | X <sup>a</sup> |
| MELD Score ≥15 | X | | |

<sup>&</sup>lt;sup>a</sup> Specifies hospitalization for ascites

The following primary efficacy assessment will be measured as an as-treated time to first occurrence of one of the following events:

#### • All-cause death

- Komodo Health: The Komodo Health data has been linked to the US National Death Index (NDI), and mortality will be recorded as date of death as recorded in the Index
- Global PBC registry: Death and date of death are reported by the physician via electronic Case Report Form (eCRF) and recorded through the CASTOR trial platform

# • Liver transplantation

- Komodo Health: The Komodo Health data will be linked to the OPTN database to ascertain whether a patient has received a liver transplant and the date of transplant.
- Global PBC registry: Liver transplant and date of transplant are reported by the physician via eCRF and recorded through the CASTOR trial platform.

# • Hospitalization for hepatic decompensation

- Komodo Health: Hospitalization for hepatic decompensation will be assessed by any hospital admission claim with the following International Classification of Diseases (ICD)-10 codes (in any position) for decompensating events
  - Variceal bleed: ICD-10: I85.01, I85.11, I86.4 and ICD-9: 456.1, 456.21, 456.8
  - Ascites: ICD-10: K70.11, K70.31, K71.51, R18.0, R18.8, J94.8, K65.2 and ICD-9: 567.23, 571.2, 789.51,789.59, 511.8, 567.23

Version 1.0: 24Jan2022

- Hepatic encephalopathy: ICD-10: B15.0, B16.0, B16.2, B17.11, B19.0, B19.11, B19.21, K70.41, K72.11, K72.90, K72.91 and ICD-9: 572.2, 070.0, 070.20, 070.41, 070.6, 070.71; or utilization of lactulose and/or rifaximin.
- Global PBC registry: Hospitalization for hepatic decompensation and date of hospitalization are reported by the physician via eCRF and recorded through the CASTOR trial platform

# 8.2. Exploratory Outcomes

There will be 3 exploratory evaluations of efficacy, measured as the as-treated:

- Time to first occurrence of all-cause death
- Time to first occurrence of liver transplant
- Time to first occurrence of hospitalization for hepatic decompensation

# 8.3. Exposure Variable

The exposure variable initiates at the OCA index date. In the Komodo database, OCA exposure will be assessed as date of first filled prescription and quantified as days supply. Discontinuation will be assessed by a gap of >90 days after previous days supply. Treatment exposure will be continued for 90 days after last days supply, after which the OCA-treated patient will be censored. In the Global PBC database, OCA exposure will be from the first physician reported utilization date to discontinuation date, plus 90 days. In this study, exposure can range from 1 to 67 months.

# 9. ASSESSMENT OF SAFETY

The objective of these replicate observational Real-world Data studies is to evaluate the effective of OCA on hepatic outcomes in patients with PBC. All patients are de-identified in the data sources. These studies are not designed to assess safety, and there are no pre-specified safety analyses. Study outcome variables collected for the 2 cohorts will be presented for analyses as aggregate data groups. The data sources will not be searched for individual patient adverse events; however, if an Investigator or Sponsor identifies adverse events that meet postmarketing reporting requirements during the course of conducting these studies, such events will be reported in accordance with applicable postmarketing reporting requirements.

# 10. STATISTICAL METHODS

# 10.1. Analysis Populations and Blinding

# 10.1.1. Analysis Populations

The statistical analysis of the HEROES PBC studies will follow a nested randomized trial emulation approach (Hernán 2008, Danaei 2013) using a treatment decision design to identify index events (Brookhart 2015). The goal of the study design is to emulate a sequence of hypothetical randomized trials. In each hypothetical trial, patients meeting the inclusion and exclusion criteria who are making the decision whether to initiate OCA-based treatment are

randomized to either continue their existing PBC treatment or switch to an OCA-based treatment. Each randomized patient is then followed until the earliest of the end of follow-up or the time of the study endpoint (death, liver transplant, or hospitalization for hepatic decompensation). Standard survival analysis methods (eg, a Kaplan-Meier estimator of the cumulative incidence function or a Cox proportional hazards model to estimate the hazard ratio) will then be used to estimate the effect of OCA on the study endpoint.

Due to the lack of randomization, non-randomized observational studies will instead be conducted, with the goal of mimicking the hypothetical randomized trial as closely as possible. All patients will be evaluated over time from the start of the study period to identify evidence of inadequate treatment response to UDCA. Each date of inadequate response identified in the data will be considered a treatment decision point, and that date will be considered an index date, with a corresponding record being created in the analytic data for that patient index. Each patient can contribute multiple index dates, and thus patient indices, corresponding to each date they have a treatment decision point, and therefore each patient may contribute person-time to multiple patient index records.

At each treatment decision point, the inclusion and exclusion criteria will be assessed (see Sections 7.2 and 7.3). For patient indices meeting the study criteria, all baseline covariates and treatment variables will be determined. Person-time corresponding to each patient index will be computed relative to the date of the index event. Notably, because prior treatment with OCA is an exclusion criterion, a patient may contribute at most one OCA-treated patient index event, though they can contribute multiple non–OCA-treated patient index events.

After the index date, follow-up will continue until the first of the composite outcome event (all-cause death, liver transplant, or hepatic decompensation), censoring, treatment discontinuation (for patient indices initiating OCA on the index date), OCA initiation (for patient indices not initiating OCA on the index date), or the end of the study period.

Because treatment will not be randomized, it is likely that OCA-treated and non–OCA-treated patient indices will differ on confounding variables, ie, variables that influence both treatment and outcome. Therefore, a simple comparison of outcomes among the OCA-treated versus non–OCA-treated patient indices is likely to yield a biased estimate of the effect of OCA on the study endpoint. To address differences in the covariate distribution between groups, the Sponsor will first conduct descriptive analyses on all baseline variables (demographics, clinical characteristics, and treatment history) for the OCA-treated and non–OCA-treated groups at index. Means, standard deviations, medians, inter-quartile ranges, and minimums and maximums will be provided for continuous variables. Counts and percentages will be provided for categorical variables. Appropriate tests comparing cohorts of interest in the primary and exploratory analyses (eg, t--test, chi-squared test) will be used based on the distribution of the measure.

Next, standardized mortality/morbidity ratio weights will be used to create a "pseudo-population" of non–OCA-treated indices with the same covariate distribution as the OCA-treated patients at the time of OCA initiation (Sato 2003), and unweighted and weighted standardized mean differences (SMDs) will be computed. SMR weights result in an average effect of treatment among the treated. They often make more efficient use of data in a situation with a small treatment group compared with inverse-probability of treatment weights. The SMR weights will be estimated as:

 $w_i^t = \frac{\hat{\pi}_i(1)}{\hat{\pi}_i(A_i)}$ , where  $w_i^t$  is the weight for patient index i,  $A_i$  is the observed level of treatment for patient index i (A = 1 if the patient index is OCA-treated, 0 otherwise),  $X_i$  is the vector of confounders measured at the index time for patient index i, and  $\pi_i(a) = \Pr(A = a | X_i)$  is the probability that patient index i receives treatment level a conditional on their covariates.

As the probabilities used to construct the weights are not known, they will be estimated using a logistic regression model. The model will be fit using observed treatment as the outcome and main effect terms for each of the covariates. Covariates (assessed in the pre-index period) will include:

- Age at index date
- Sex
- Most recent liver biochemistry levels (TB, ALP, ALT, AST)
- Most recent platelet counts
- Time (in months) since UDCA failure
- Clinical evidence of portal hypertension (platelets <150,000 and/or non-bleeding varices)
- Cirrhosis
  - Komodo Health: cirrhosis diagnosis with liver imaging and/or biopsy within 6 months before diagnosis
  - Global PBC registry: biopsy stage 4, transient elastography ≥16.9 kPa, radiological evidence (nodular liver or enlargement of portal vein with splenomegaly), clinical features of portal hypertension defined as platelet count <140 000/mm³ with persistent decrease in serum albumin; or, TB >2x ULN, or prothrombin time/INR > ULN (not due to antithrombotic use)
- Most recent Charlson Comorbidity Index Score (Glasheen 2019)
- Insurance type at the index date (Komodo Health only: commercial, Medicare, Medicaid, dual eligible, other)

All diagnosis, procedure and laboratory codes used to define the control variables are listed in Appendix A.

Once the weights are constructed, a table of weighted SMDs between the groups will be constructed to assess balance. An absolute SMD of greater than 0.1 will indicate potentially problematic residual imbalance for the particular covariate. In the case that either the model-fitting algorithm fails to converge, or residual imbalance exists after weighting, the study team will attempt to reduce model complexity or reduce imbalances by implementing one or more of the following actions:

- Adding/removing interaction terms (1st order or higher)
- Using a spline for continuous variables
- Shrinking all coefficients in the model using a penalty

To protect the integrity of the research results, all decisions about updating the analysis will be made by the Investigators without knowledge of how those decisions might affect the outcome (Clean Room Committee [CRC], see Section 10.11). Each decision for a set of actions will be tracked in a study log along with the results presented to the analysis team to inform the action. The final weights will be used for the main analysis. Results for each stage of the developed weights will be documented and presented as supplementary material (and decisions will be recorded in the study log).

Under the identification conditions of causal consistency (Cole 2009, VanderWeele 2009, Pearl 2010), (partial) conditional exchangeability (Greenland 1986, Sarvet 2020), and positivity (Westreich 2010, Petersen 2012), the pseudo-population resulting from weighting the person-indices will emulate the data (at baseline) of the aforementioned hypothetical randomized trial.

# **10.1.2. Blinding**

To ensure that knowledge of outcomes does not influence group creation, all persons involved in the studies will be kept blind to outcomes (death, liver transplant, hospitalization for decompensation) until after the analytic groups are created and the SMR weights are finalized. The event file will be kept separate from the primary data containing patient demographic, medical history, treatment, and laboratory data and will not be accessible to study personnel. Once the OCA-treated and non–OCA-treated datasets are created and approved by the CRC, the CRC will notify non–study-affiliated designees at each site that the event data can now be accessed in order to perform the effect size analysis and statistical testing.

# 10.2. Estimation of Effect Size

The causal effect of OCA-containing treatments versus non–OCA-containing treatments on the study endpoints will be quantified using a hazard ratio. The hazard ratio will be estimated using a weighted version of the sequential Cox proportional hazards model (Gran 2010). This approach entails fitting a weighted Cox proportional hazards regression to the person-index dataset, with weights created as previously described, treatment included as a non–time-varying indicator of baseline treatment, and the timescale being specified as time since the index event. In addition to adjusting for confounding via SMR weighting, baseline covariates for each person-index will also be included in the regression model to address possible informative censoring by baseline variables. To test for heterogeneity of effects across each of the nested 'trials', an interaction term between treatment and an indicator representing each trial will be included in the model. A non-significant coefficient for the interaction variables will indicate heterogeneity.

In randomized trials, a common approach to address imperfect treatment adherence is to censor patients when they deviate from their assigned treatment, a so-called per-protocol analysis (Hernán 2017). An analogous approach can be used for non-randomized observational studies. Here, a person-index is censored when they deviate from their initial treatment. For instance, if a person-index received non-OCA treatment at baseline but OCA was initiated 6 months after the index date, that person-index would be censored at 6 months. Similarly, if a person-index received OCA at baseline but discontinued OCA, that person-index would be censored once the definition of OCA discontinuation is met, with an extension of 3 months after that time to allow

for duration of effect after discontinuation. As a result of this artificial censoring, all person-time included in the analysis reflects adherence to initial treatment. Similarly, by excluding person-time occurring after loss to follow-up, all included person-time additionally reflects remaining time under study.

Because treatment non-adherence and loss to follow-up may not occur completely at random, those who remain uncensored may differ from the overall study population on key prognostic factors. To address these differences, the Sponsor will include baseline covariates in the Cox model that are potential predictors of both the study outcomes and censoring.

# 10.3. Hypotheses

# 10.3.1. Primary Hypothesis

These studies are intended to assess whether there is a difference between patients treated with OCA and comparable OCA-eligible patients who are not treated with OCA in the time from index to the first occurrence of all-cause death, liver transplant, or hospitalization for hepatic decompensation.

Two-sided hypotheses are expressed in terms of:

- The null hypotheses (H<sub>0</sub>) that the 2 hazard functions are the same, as determined by a hazard ratio (HR) equal to 1; that is, at every timepoint, the instantaneous event rates are the same for the OCA and control populations.
- The alternative hypothesis (H<sub>1</sub>) that the 2 hazard rates are not the same ( $HR \neq 1$ ).

# **10.4.** Determination of Sample Size

Using the sample size in the 2 populations (Section 6.2), the Sponsor computed power to detect treatment effects (relative hazards) of varying sizes, estimated using Cox proportional hazards regression. Computations are based on the formulae of Schoenfeld 1983. To account for confounding control due to the application of IP weights, the Sponsor inflated the variance from the Schoenfeld formula using factors derived by Shook-Sa 2020. It was conservatively assumed just one control observation per patient. In the Komodo Health data, a preliminary investigation found that approximately 395 patients who meet entry criteria will initiate OCA and that 5916 patients will contribute at least one record to the control group (UDCA nonresponders). In the Global PBC registry, the Sponsor expects to have 344 patients meeting entry criteria who initiate OCA, and 2200 who contribute at least one observation to the control group. Power in both cohorts was computed for relative hazards ranging from 0.5 to 0.9 with an alpha level of 0.05. The Sponsor considered baseline event rates during follow-up from 5% to 15% and variance inflation corresponding to mild confounding (VIF=1.05), moderate confounding (VIF=1.5), and strong confounding (VIF=2.0). In each study, power was plotted under these assumptions against a reference line of 80% power under moderate confounding (VIF=1.5) (Figure 2).

Under mild confounding, both studies will be well-powered to detect an HR of 0.5. For moderate confounding, the Komodo Health study will be adequately powered to detect HR of 0.5 for event rates >6%. The Global PBC registry will be adequately powered to detect event rates >8%. Under strong confounding, the Komodo Health study will be adequately powered to detect

HR of 0.5 for event rates >9%. The Global PBC registry will be adequately powered to detect event rates >11%. Power decreases for more moderate HRs. None of the studies under even the most favorable assumptions will be able to detect HRs of 0.9. The Sponsor notes that the assumptions made here are conservative; in particular, it is expected that many more than one control observation and that the addition of lab data from LabCorp (as noted in Section 6.2) will substantially increase the size of both groups in the Komodo Health study.

Figure 2: Power estimates by Hazard Ratio by Level of Confounding for Komodo Health (A) and Global PBC Registry (B).



# 10.5. Primary Efficacy Analysis

Standard error estimation will proceed using the nonparametric cluster bootstrap (Davison 2013) as has been suggested for nested trial designs using Cox proportional hazards regression (Gran 2010). The standard error will be used to calculate the 95% CI of the hazard ratio and to conduct statistical hypothesis testing. A total of 1000 bootstrap replicates will be used. Bootstrap sampling will occur at the patient level, rather than the patient index level, thus preserving the covariance structure between patient indices and properly accounting for variance inflation due to the covariance between analytic units. Within each bootstrap replicate, all aspects of estimation will be repeated, including the fitting of the treatment model, the construction of the weights, and the fitting of the weighted Cox proportional hazards model used to estimate the treatment effect. The standard deviation of the bootstrap estimates of the treatment effect will be used as an estimate of the standard error. A Wald test will then be conducted using the bootstrap standard error (Cameron 2008). The test statistic is defined as

 $w = \frac{\hat{\beta}}{s_{\hat{\beta}}}$ , where  $\hat{\beta}$  is the estimated coefficient of OCA treatment from the fitted Cox model and  $s_{\hat{\beta}}$  is the bootstrap standard error of the estimated coefficient. With a sufficient sample size, w will follow a standard normal distribution and the p-value will be computed as the probability of a normal random variable being greater than |w| or less than -|w|. A p-value less than 0.05 will be considered statistically significant.

# 10.6. Exploratory Analyses

Each component of the study endpoint (all-cause death, liver transplant, and hospitalization for hepatic decompensation) will be assessed separately. For the outcome of death, the analysis will proceed using the same approach as for the primary effect size estimation. For the outcome of liver transplant, death will be treated as a competing event. Here, follow-up will end at the earliest of the end of follow-up, liver transplant, death, or censoring. The analysis will proceed as previously described, but instead of a Cox proportional hazards model, a Fine-Gray proportional subdistribution hazards model will be used (Fine 1999). Similarly, for the outcome of hospitalization for hepatic decompensation, death and liver transplant will be treated as competing events.

# 10.7. Handling of Dropouts or Missing Data

Patients who disenroll from the covered health plans in Komodo Health or from the Global PBC registry are right-censored at time of disenrollment.

Dropout / disenrollment will be assumed to be uninformative conditional on the included baseline covariates in the Cox model (see Section 10.2). Missing baseline data will be assumed missing completely at random, and a complete case analysis (listwise deletion) will be conducted. During the conduct of the studies, the CRC may recommend refining the missing data strategy to better address any observed pattern of missing data.

# 10.8. Subgroup Analyses

The entire analysis will be repeated separately by patient race (Komodo Health only), age (categorical), sex, region, absence/presence of cirrhosis, and pre-/post-COVID. Because race is not completely captured in Komodo Health, these analyses will only include those with non-missing values for race.

# 10.9. Sensitivity Analyses

A quantitative bias analysis will be used to assess the sensitivity of the estimates to violations of the assumption of no unmeasured confounding. To conduct this analysis, it will be assumed that the hazard ratio is a reasonable approximation of the odds ratio, and then previously published formulas for the relation of unadjusted or partially adjusted to adjusted odds ratios will be used to estimate the effect, given inputs for the strength of the confounder treatment and confounder outcome relationships (Lash 2021). The analysis will be conducted across a range of values for the input parameters to assess how much the effect changes given different confounder relationships. Specifically, given the (adjusted for known confounders) odds ratio for the association between the unmeasured confounder and the outcome  $(OR_{DZ})$  and the prevalence of the confounder among the OCA-treated  $(P_{Z1})$  and non-OCA-treated  $(P_{Z0})$  (each assumed

homogeneous across levels of known confounders), the relationship between the partially adjusted and fully adjusted odds ratios is  $\frac{OR_{partial}}{OR_{full}} = \frac{OR_{DZ}P_{Z_1} + 1 - P_{Z_1}}{OR_{DZ}P_{Z_0} + 1 - P_{Z_0}}.$ 

# 10.10. Assessment of Claims-based PBC Definition

The Komodo Health data are claims-based. Per AASLD guidelines, PBC diagnosis is based on the presence of  $\geq 2$  of 3 diagnostic factors:

- History of elevated ALP levels for at least 6 months
- Positive AMA titer
- Liver biopsy finding consistent with PBC

AMA is normally assessed once to diagnose PBC, and the test may have occurred years prior to entry into the Komodo Health claims database. Indeed, a preliminary analysis shows that ~10% of patients with a PBC diagnostic code have an AMA test result in the database. As AMA cannot be used in the definition of PBC, a claims-based analysis will be used to identify PBC patients in claims data requiring 2 outpatient claims or 1 inpatient claim based upon the work of Meyers (Meyers 2010).

Using Canadian ambulatory care and inpatient records, Meyers found that a 2-outpatient claim algorithm had 89% positive predictive value (PPV) when compared to AMA-verified definite, probable, or suspected PBC. A single inpatient claim had 81% PPV, with limited incremental benefit of 2 claims (86% PPV).

In these studies, in addition to the claims criteria, evidence of UDCA use is required, which the Sponsor believes will further improve the PPV of the claims-based algorithm. To validate this approach, the Sponsor will conduct sensitivity and specificity analyses using AMA as the gold standard of PBC diagnosis within the Komodo Health database. The subpopulation of patients with AMA test results (positive vs negative) will be compared to those with a positive and negative diagnosis by the claims + UDCA definition. The sensitivity of the non–AMA-based definition will be defined as the proportion of patients classified as having PBC with the gold standard definition who are also classified as having PBC with the non–AMA-based definition. The negative predictive value of the non–AMA-based definition will be defined as the proportion of patients not classified as having PBC with the non–AMA-based definition who are also not classified as having PBC with the gold standard definition. The specificity and PPV will be assumed to be equal to 1, as the non–AMA-based definition will capture a subset of those individuals classified as having PBC by the gold standard definition.

# 10.11. Clean Room Committee

In studies of existing data, decisions about study design or analysis should not be informed by knowledge of how such decisions might affect study results. The study team has attempted to pre-specify all statistical analysis plans to a sufficient degree of detail that ambiguity about how the results will be obtained is minimized. However, often data will need to be examined to inform key aspects of the study design or analysis, and in other cases, issues discovered during analysis might require certain deviations from the planned design and/or analysis.
To avoid biasing point estimates and standard errors for the primary comparative analysis, the individuals making these decisions will be isolated from knowledge about how these decisions might affect outcomes. To do this, the 3 individuals will be designated to be members of the CRC, and this designation will be recorded in the study log. Analysts will have direct access to the data and will build all analytic files and implement all data analysis. Study team members not designated as CRC members will work with the analysts to review and understand output tables.

Members of the CRC will make all decisions about the conduct of these studies, including decisions about protocol deviations as well as the reporting and interpretation of results in reports. Additionally, based on data supplied to them by the analysts, the CRC will make decisions about changes in analytic approaches, model specification, group inclusion/exclusion criteria, and variable definitions. The data supplied by the analyst should not provide any direct information about how such protocol changes might affect results. To accomplish this, preliminary results that contain outcome statistics summarized by group (OCA-treated versus not OCA-treated) will not be presented to the Investigators. If, for some reason, results need to be presented by group, the group will be masked by the analysts. All aspects of this process will be tracked, specifically:

- All requests for interim data or results will be entered into the study log where they can be viewed by all study team members.
- All protocol deviations will be logged along with the rationale for the change. Protocol changes will not be made unless all Investigators agree to the change.
- Minutes of meetings in which decisions about protocol changes are made will be saved.
- The original protocol as well as all modified versions will be accessible to all Investigators and analysts.

The original protocol and the study log will be made available as appendix material for all reports and publications.

## 11. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

The data in these studies are de-identified. The Komodo Health data use agreements and the Global PBC registry Institutional Review Board (IRB) approval specify that these data may not be re-identified. In addition, the Global PBC registry site agreements do not allow for the transfer of data outside of the Global PBC registry.

The Clinical Research Organization (CRO) will ensure the Investigator's understanding of all applicable regulations and standard operating procedures (SOPs) and will ensure an understanding of the protocol and maintenance of all requisite documentation. The CRO will have full access to the Komodo Health data and analyses to be able to ensure these studies are conducted per protocol. The CRO can also review data and programming on site with a member of the Global PBC Study Group.

A Study Data Tabulation Model (SDTM) dataset will be provided to the FDA for the Komodo Health dataset. Should the FDA have questions or queries, a member of the Global PBC Study

Group will make themselves available on site at the FDA with a laptop computer containing the Global PBC registry analytic dataset and can both review data and run queries as required by the FDA.

# 12. QUALITY CONTROL AND QUALITY ASSURANCE

In 2021, the FDA released 4 draft guidance documents defining data quality, management, and analyses of real-world data, including guidance specific to claims data and disease registries. Given the extensive documentation requirements, separate supplemental protocols will be submitted, one for the Global PBC registry and one for the Komodo Health dataset.

## 12.1. Data Collection and Transfer

#### 12.1.1. Komodo Health

Komodo Health merges administrative claims across >350 health plans including commercial (63%); Medicaid (23%); Medicare (10%); dual eligible (<1%); and other (2%). The dataset represents more than 325 million unique patients in the US between June 2015 and July 2021. The datasets include all inpatient, outpatient, and procedure claims, as well as service dates, associated ICD-9 and ICD-10 codes, and provider data.

Data from each payer are tokenized, deidentified, and encrypted by the individual payer (see Section 12.2.2). Some examples of file formats Komodo Health intakes from sources include TXT, CSV, and DAT file types. Komodo Health commonly receives data as (but not limited to) comma-delimited, pipe-delimited, and tab-delimited files. A transit token specific to the payer and Komodo Health is used, and once received the data are de-encrypted, including a final patient token. Thirty-six percent of plans transfer their data through a Komodo Health secure FTP site; 64% of plans provide a secure FTP site to Komodo Health to retrieve the data. Komodo Health receives and stores data in AWS S3 buckets.

Plans provide uncurated (raw) data. Data cleaning, such as deduplication, will be specified in the supplemental submission. Cleaned data are merged and linked via token, thus patients are able to be followed longitudinally across plans that contribute data. After Komodo Health finishes processing the data, they are made available as a Snowflake database in the Sentinel cloud environment.

## 12.1.2. Global PBC Registry

Data for the Global PBC registry is collected through the CASTOR trial platform. The CASTOR System, which has been employed for registrational trials, includes eCRFs, cloud-based data collection, and download of data in SAS format for analysis. The data are only transferred to the University Health Network system, with no additional data transfer, and are analyzed in the SAS environment. The eCRF prevents the input of test values outside of medically plausible range and the input of duplicate data. Source data cannot be modified. The Global PBC registry protocol, eCRFs, and all data cleaning and transformations of variables included in this analysis will be specified in the supplemental submission.

#### 12.1.3. National Death Index

The NDI is a central computerized index of death record information on file in state vital statistics offices. The Centers for Disease Control and Prevention and the National Center for Health Statistics compile deaths annually from computer files submitted by state vital statistics offices. Numerous studies have confirmed the validity of the NDI. The NDI has previously been linked to the Komodo Health database (see Section 12.3) and the datafile will be kept firewalled from analysts until the CRC authorizes unblinding. The NDI will be used to ascertain death as part of the composite endpoint.

The Komodo Health data contains information on hospital discharge status, including death at discharge. Death status, combined with a lack of addition claims >30 days after deaths will be compared to the NDI database. If a death on hospital discharge (plus lack of additional claims) is observed in the Komodo database but not in the NDI database, it will be included as a primary endpoint.

## 12.1.4. Quest Diagnostics

Quest Diagnostics has >2000 testing facilities with specimens processed at 26 central laboratories in the US (excluding those devoted exclusively to clinical trials). Specimen collection and testing protocols are standardized nationally. Date of test, laboratory value results, normal range limits, and associated ICD-10 codes are entered at each lab facility. Data are sent electronically to the testing site, and also to a centralized main frame and entered into the national database within 7 days. Specifications on data storage, transfer, and cleaning will be included in a supplemental submission.

These studies will utilize ALP, TB, ALT, AST, and platelets to propensity weight treated and untreated patients at index, and to determine UDCA treatment failure. AMA data will be used to validate the ICD-10 PBC claims diagnostic criteria.

#### **12.1.5.** LabCorp

LabCorp has >2100 testing facilities with specimens processed at 15 primary laboratories in the US (excluding specialty testing facilities such as oncology and genetic testing). Specimen collection and testing protocols are standardized nationally. Date of test, lab value results, normal range limits, and associated ICD-10 codes are entered at each lab facility. Data are sent electronically to the testing site, and also to a centralized main frame and entered into the national database. Specifications on data storage, transfer, and cleaning will be included in a supplemental submission.

These studies will utilize ALP, TB, ALT, AST, and platelets to propensity weight treated and untreated patients at index, and to determine UDCA treatment failure. AMA data will be used to validate the ICD-10 PBC claims diagnostic criteria.

## 12.1.6. OPTN Transplant Registry

OPTN collects and reports data on every US organ donor, transplant candidate, recipient, and outcome. Data are collected through a standardized eCRF using the online UNet database system. Specifications on data storage, transfer, and cleaning will be included in a supplemental submission.

The OPTN registry will be the primary data source to ascertain liver transplant as part of the composite endpoint. The Komodo Health data contains information on hospital admissions, including codes for liver transplant (see Appendix A). Hospitalization for liver transplant in Komodo Health claims will be compared to the OPTN database. If a liver transplant is recorded on hospital discharge but not in the OPTN database, it will be included as a primary endpoint.

## 12.2. Data De-identification

## 12.2.1. Global PBC Registry

The data collected at each site are de-identified by removing all identifying data fields (name, address, date of birth, etc.) prior to being sent to the Central Coordinating Site. A unique Global PBC Study Group study number is assigned to each site and each participant within the site and does not utilize identifying information in creating the patient number. Identifiers and their relation to the Global PBC Study Group number are maintained only at the study site and not by the central Data Coordinating Site.

#### 12.2.2. Komodo Health

Datavant's de-identification engine is designed for use on structured healthcare data. The de-identification program performs 2 functions: de-identification of the data set through removal or modification of identifying data, and the insertion of encrypted patient tokens. De-identification includes the following:

- Zip Code: Reduced to the initial three characters to define a zip area. Based on the Health Insurance Portability and Accountability Act (HIPAA) rules, however, even three-digit zip areas with a combined population of less than 20,000 are either nulled out or are combined again with additional zip zones to ensure that populations exceed this minimum.
- Date of Service: Dates of service (eg, admission dates, discharge dates, prescription fill dates, and procedure dates) are typically preserved when using a statistical de-identification methodology.
- Date of Birth: Converts all birth dates to birth year. All dates of birth where the individual aged ≥89 years as of the date of de-identification would be modified to reflect an age of 89.
- Medical Records Numbers: Removed where present
- Telephone Numbers: Removed where present
- Email Address: Removed where present
- Social Security Numbers: Removed where present
- Beneficiary Numbers: Removed where present
- Vehicle Information: Removed where present
- Device Identifiers and Serial Numbers: Removed where present
- URL Addresses: Removed where present

- IP Addresses: Removed where present
- Biometric Values: Removed where present in claims data; retained in Quest Diagnostics and LabCorp
- Image Fields: Removed as defined by the data source

Datavant does not perform de-identification and tokenization itself and does not have access to the user's system or identifying information. The de-identification process is executed by the institution that owns the data, ie, Datavant's technology is installed and run locally behind the users' firewalls.

# 12.3. Data Linkages

Two sets of linkages are relevant for Komodo Health: initial link of contributing administrative claims databases; and linkage of laboratory data (LabCorp and Quest Diagnostics), death date (NDI), and transplant date (OPTN registry). All data linkages will be done through Datavant tokenization.

Across all datasets, as the Datavant program de-identifies a patient record, it also generates one or more tokens for that record. Tokens are based on the personally identifying data in the record, but the token itself does not incorporate this information in the identifier. The tokens are consistently created from any data set where the underlying identifying information is the same. Matching tokens are used to link a patient's record in one data set with a record for the same patient in a different set, without exposing the identifying information of that patient. Matching can be deterministic (eg, based on social security number) or probabilistic (eg, based on combination or name, sex, birthdate, 3-digit zip code, etc).

The tokens used to link records in de-identified data sets cannot be reversed to reveal the patient's identifying information. The first step of the token creation process is the use of an irreversible hash function, which ensures that the patient's personally identifying information used to create the token cannot be recovered from the output value. In the second step of the process, the hash value (ie, "Master Token") is encrypted with a site-specific encryption key to generate the final encrypted patient token. While the same patient information will always create the same Master Token, site-specific encryption means that a single patient will have a unique token (ie, a "site-specific token") in each specific user's data set. Site-specific encryption ensures that a breach at one data site will never compromise the tokens or protected health information at any other data site. Datavant's QA testing protocols and results will be included in the supplementary submission.

Across all datasets, Datavant will create 2 tokens based on:

- Last name + first name + gender + date of birth
- Last name (soundex) + first name (soundex) + gender + date of birth

In the event this produces 2 patients with one token (called a "collision") or one patient with 2 tokens, Datavant will then match on social security number and/or address (when available in the dataset). In the overall Komodo Health claims database, in the match with the NDI, and in the match with Quest Diagnostics data, this has produced 99% exact match. In the subset of

PBC patients, only 873 of 164,942 patients are flagged as a collision and have been removed from analysis. The same process will be used with the OPTN transplant data.

## 12.4. Data Harmonization

The Global PBC registry collects data via a standardized eCRF. As such, data harmonization across data sources is not required.

The Komodo Health database merges administrative claims data from multiple insurers in the US. Claims are then merged with NDI for date of death; LabCorp and Quest Diagnostics databases for laboratory tests and values; and OPTN transplant registry for date of liver transplant. Below are the data sources and variables for which data harmonization is required and performed.

#### 12.4.1. Komodo Health and National Death Index

The primary endpoint is a composite of all-cause death, liver transplant, and hospitalization for hepatic decompensation. The primary source for death will be the NDI. The Komodo Health claims database contains hospital discharge status, including "death." Hospital discharge of death will be compared to the NDI. Should a death be recorded on hospital discharge but not in the NDI, and if the patient has no healthcare claims 30 days after the "death" discharge, the patient will be coded as a death using the hospital discharge date.

## 12.4.2. Komodo Health and OPTN Liver Transplant

The primary endpoint is a composite of all-cause death, liver transplant, and hospitalization for hepatic decompensation. The primary source for liver transplant will be the OPTN transplant registry. Hospitalization for liver transplant in Komodo Health claims also will be ascertained through inpatient ICD-10 codes (see Section 12.4.3 and Appendix A). Komodo Health liver transplant claims will be compared to the OPTN database. Should a liver transplant be recorded for a hospitalization but not in the OPTN database, it will be included as a primary endpoint.

# 12.4.3. Komodo Health Hospitalization for Hepatic Decompensation

The primary endpoint is a composite of all-cause death, liver transplant, and hospitalization for hepatic decompensation. The primary source for hospitalization for hepatic decompensation will be Komodo Health claims. The definition will include inpatient admission ICD-10 codes that appear in any position, and includes:

- Variceal bleed: ICD-10: I85.01, I85.11, I86.4 and ICD-9: 456.1, 456.21, 456.8
- <u>Ascites</u>: ICD-10: K70.11, K70.31, K71.51, R18.0, R18.8, J94.8, K65.2 and ICD-9: 567.23, 571.2, 789.51,789.59, 511.8, 567.23
- <u>Hepatic encephalopathy</u>: ICD-10: B15.0, B16.0, B16.2, B17.11, B19.0, B19.11, B19.21, K70.41, K72.11, K72.90, K72.91 and ICD-9: 572.2, 070.0, 070.20, 070.41, 070.6, 070.71; or utilization of lactulose and/or rifaximin

As ICD-10 codes are standard across the US healthcare industry, there is no need for further harmonization across contributing health plans.

## 12.4.4. Quest Diagnostics and LabCorp

Within each laboratory provider, sample collection, test, and normal ranges are standardized. Collection and transport specifications, laboratory method, and normal ranges for each test are provided by each lab below.

- Total bilirubin (test code: Quest 285, LabCorp 001099)
  - Quest Diagnostics: Samples are collected in sodium heparin (green-top) or lithium heparin (green-top) tubes, spun in a serum separator tube, transported in a serum separator tube wrapped in foil or transferred to an amber transport vial, and stored/transported at room temperature with stability up to 24 hours.
     Spectrophotometry is performed on 1 mL serum. ULN is 1.2 mg/dL.
  - LabCorp: Samples are collected in red top gel-barrier tube or lithium heparin (green-top) tubes, with serum separation in ≤45 minutes, and stored/transported at room temperature with stability up to 3 days. Spectrophotometry testing is performed on 1 mL serum. ULN is 1.2 mg/dL for ≥18-year-olds.
- Alkaline phosphatase (test code: Quest 234, LabCorp 001107)
  - Quest Diagnostics: Samples are collected in sodium heparin (green-top) or lithium heparin (green-top) tubes, spun and transported in a serum separator tube, and stored/transported at room temperature with stability up to 7 days.
     Spectrophotometry is performed on 1 mL serum. ULN in U/L for 18- to 19-year-olds is 169 for men and 128 for women; for 20- to 49-year-olds is 130 for men and 125 for women; and for ≥50-year-olds 144 for men and 153 for women.
  - LabCorp: Samples are collected in red top gel-barrier tube or lithium heparin (green-top) tubes, with serum separation in ≤45 minutes, and 1 mL serum transported in plastic separator tube, and stored/transported at room temperature with stability up to 14 days. Kinetic testing is performed on 1 mL serum. ULN in IU/L for 18- to 20-year-olds is 125 for men and 106 for women; for ≥21-year-olds is 121 for men and women.
- Alanine aminotransferase (test code: Quest 823, LabCorp 001545)
  - Quest: Samples are collected in sodium heparin (green-top) or lithium heparin (green-top) tubes, spun and transported in a serum separator tube, and stored/transported at room temperature with stability up to 72 hours.
     Spectrophotometry is performed on 1 mL serum. ULN in U/L for 18- to 19-year-olds is 46 for men and 32 for women; for ≥20-year-olds is 46 for men and 29 for women.
  - LabCorp: Samples are collected in red top gel-barrier tube or lithium heparin (green-top) tubes, with serum separation in ≤45 minutes, and stored/transported at room temperature with stability up to 7 days. Kinetic testing is performed on 1 mL serum. ULN is 44 IU/L for ≥18-year-olds.

• Aspartate Aminotransferase (test code: Quest 822, LabCorp 001123)

Quest Diagnostics: Samples are collected in sodium heparin (green-top) or lithium heparin (green-top) tubes, spun and transported in a serum separator tube, and stored/transported at room temperature with stability up to 4 days.
 Spectrophotometry is performed on 1 mL serum. ULN in U/L for 18- to 19-year-old men and women is 32; for men, 20- to 49-year-olds is 40 and >50-year-olds is 35; for women, 20- to 44-year olds is 30 and >45-year-olds is 35.

- LabCorp: Samples are collected in red top gel-barrier tube or lithium heparin (green-top) tubes, with serum separation in ≤45 minutes, and stored/transported at room temperature with stability up to 7 days. Kinetic testing is performed on 1 mL serum. ULN is 40 IU/L for >18-year-olds.
- Platelets (test code: Quest 723, LabCorp 005249)
  - Quest Diagnostics: Samples are collected in lavender-top (EDTA) tubes and stored/transported at room temperature with stability up to 48 hours. Testing is performed on 0.5 mL whole blood using an automated cell counter. Lower limit of normal (LLN) is 150,000 per uL for ≥18-year-olds.
  - LabCorp: Samples are collected in lavender-top (EDTA) tubes, immediately inverted 8 to 10 times, and stored/transported at room temperature with stability up to 1 day. Testing is performed on 0.5 mL whole blood using an automated cell counter. LLN is 150,000 per uL for ≥18-year-olds.

#### 12.4.5. Cirrhosis

In the Global PBC registry, cirrhosis is assessed as positive for one or more of the following criteria:

- Biopsy Stage 4;
- Transient elastography ≥16.9 kPa;
- Radiological evidence (nodular liver or enlargement of portal vein + splenomegaly);
- Clinical features of portal hypertension defined as platelet count <140 000/mm³ with: persistent decrease in serum albumin; or, TB >2x ULN; or prothrombin time/INR > ULN (not due to antithrombotic use)

In the Komodo Health database, imaging data are not available and measures such as INR are not consistently collected. The Sponsor created and validated an algorithm for a claims-based cirrhosis diagnosis, defined as: cirrhosis ICD-10 (K74.5; K74.60; K74.69) with liver imaging and/or biopsy in 6 months preceding diagnosis (for imaging codes see Appendix A). Prevalence estimates in patients with PBC based on these codes in the HealthCore and Optum databases, stratified by decompensation and portal hypertension, were compared to data from the Global PBC registry (Table 2). As shown, the concordance was high. Additional analyses examining the association between these groups and clinical outcomes (death, liver transplant and hepatic decompensation) demonstrated that the expected relationships, with cirrhosis in the presence of portal hypertension or decompensation significantly increasing risk of death, liver failure and liver transplantation (Figure 3).

Table 2: Comparison of Imaging-based (Global PBC) and Claims-based (HealthCore, Optum) Prevalence of Cirrhosis in PBC Patients.

| | Global PBC | Optum | HealthCore |
|---|---|---|---|
| PBC | N=2,982 (100%) | N=4,328 (100%) | N=4,348 (100%) |
| Compensated non-cirrhosis | N=2,275 (76.3%) | N=3,303 (76.3%) | N=3,317 (76.3%) |
| Compensated cirrhosis, without portal hypertension | N=314 (10.5%) | N=271 (6.3%) | N=225 (5.2%) |
| Compensated cirrhosis, with portal hypertension | N=105 (3.5%) | N= 276 (6.4%) | N=295 (6.8%) |
| Decompensated | N=283 (9.5%) | N=478 (11.0%) | N=511 (11.8%) |

Figure 3: Incidence Rates for Major Hepatic Events Stratified by Cirrhosis, Portal Hypertension and Hepatic Decompensation in the Optum (A) and HealthCore (B) Databases



## 12.5. Characterization of Missing Data

Missing data will be assumed to be missing at random. As per FDA draft real-world evidence (RWE) guidelines, missing data are characterized by year (see Appendix B) and will undertake an analysis of secular trend to determine if missingness varies by time. Should secular trends exist, the CRC will determine the best approach to addressing bias, and that approach will be included in a protocol revision.

# 12.6. Data Management and Analysis SOPs

The FDA draft guidance on RWE requires a data management plan as well as copies of all relevant data management and analysis SOPs. These will be included in a supplemental submission and defined separately for the Global PBC study group and the CRO analyzing the Komodo data.

# 12.7. Audits and Inspections

The Investigators should understand that it may be necessary for the Sponsor, the IRB/Independent Ethics Committee (IEC), and/or regulatory agencies to conduct one or more site audits during or after the study and agree to allow access to all study-related documentation and information and be available for discussion about the study.

# 12.8. Quality Control and Quality Assurance

Logic and consistency checks will be performed on all data in the database to ensure accuracy and completeness. SOPs from the CRO analyzing the Komodo data and the Global PBC Study Group governing data management and analysis will be provided in a supplemental submission.

Given the short length of the study conduct period (approximately 6 months for analysis and clinical study report), the Sponsor will conduct a single monitoring visit at each site. Study records will be reviewed to ensure maintenance and documentation of complete, accurate, legible, well-organized, and easily retrievable data. The Sponsor will ensure the Investigator's understanding of the protocol, reporting responsibilities, and the validity of the data. This will include ensuring that full and appropriate essential documentation is available. To perform analytic file and analysis verification, the Sponsor must be given access to the analytic file, SAS code and code annotation. The Sponsor will not alter data or programming, nor will transport any data from the site.

# 12.9. Data Retention and Archiving Study Documents

The CRO analyzing the Komodo data and the Global PBC Study Group will retain the data and all study documents after delivery of the project for a maximum period as required by the applicable regulatory requirement(s) or the Sponsor. In the event that storage of data becomes a problem at any time during this period, the Sponsor should be consulted for assistance. At the end of the minimum period, the CRO and the Global PBC Study Group should obtain written authorization from the Sponsor before the destruction of any records. The Sponsor will inform the CRO and the Global PBC Study Group should it become aware of any changes in storage requirements.

## 13. PROTECTION OF HUMAN SUBJECTS

These studies will be conducted in accordance with HIPAA regulations and US standards of privacy of individually identifiable health information.

The Global PBC registry was approved by the University Health Network IRB at the University of Toronto (CAPCR ID: 19-5678).

All data used in these studies are anonymized, and analyses will be performed on de-identified patient-level datasets. While patient data will be anonymized and the studies are observational and retrospective in nature and thus would qualify for exemption under the Common Rule, these studies are being submitted to Western IRB for full review.

The data system will be maintained and secured as requested by the US patient privacy regulations. Processes assuring data security will be employed during data extraction, storage, and backup. The data and all study documents will be kept until the Sponsor's written notification that records may be destroyed.

#### 14. ADVERSE EVENT REPORTING

As stated in Section 9 (Assessment of Safety), these studies are not designed to assess safety. Study outcome variables collected for the 2 cohorts will be presented for analyses as aggregate data groups. The data sources will not be searched for individual patient adverse events. However, if an Investigator or the Sponsor identifies adverse events that meet postmarketing reporting requirements during the course of conducting these studies, such events will be reported in accordance with applicable postmarketing reporting requirements.

#### 15. PUBLICATION POLICY

The Sponsor intends to publish the results of all of the studies that it sponsors, regardless of outcome and consistent with the Declaration of Helsinki. Consistent with the recommendations of the editors of several leading medical journals, the International Committee of Medical Journal Editors (ICMJE), authorship of publications resulting from Intercept-sponsored studies should fairly recognize the activities of those that have made a significant contribution to the study (http://www.icmje.org). Thus, it is anticipated that authorship will reflect the contribution made by the Sponsor personnel, the Investigators, and others involved, such as statisticians.

In recent years, issues about conflicts of interest and accuracy of study data have been raised in the medical press. Accordingly, the Sponsor has developed publication guidelines for studies that are appropriate for these studies. Key issues include the following:

- Clinical Trial Registries (eg, www.clinicaltrials.gov, www.clinicaltrialsregister.eu): A description of these studies and relevant design elements (eg, basic design, objectives and endpoints, sample size, study population, and key inclusion/exclusion criteria) and results will be published online in a manner consistent with applicable regulatory guidelines.
- Overview: Investigators, reviewers, and editors will have the right to audit the data to verify its accuracy.

• Responsibility: Each Investigator is responsible for the accuracy and completeness of all data from her/his site. The Sponsor (or its representatives) is responsible for the accuracy of the data entered into the study databases and the analyses conducted.

- Authorship: Intercept, in collaboration with the Investigators, will establish the appropriate authorship and responsibility for drafting study documents in accordance with the principles of the ICMJE. All manuscripts will be reviewed and agreed upon before submission for publication by all authors.
- Intercept Review of External Manuscripts: Investigators must submit any drafts of any publications or presentations that may arise from these studies to the Sponsor for review and approval and to ensure consistency with the policy in this protocol at least 30 days prior to submission for publication or presentation. The Sponsor will have the right to request appropriate modification to correct facts and to represent its, or the Publication Committee's, opinion if these differ with the proposed publication.
- Confidentiality: Investigators will conduct all interactions with the company and with third parties consistent with the executed confidentiality agreements. While publication, by intention, presents the critical scientific data in a public forum, some information (such as future plans, results of preclinical studies, or chemical formulae) may still need to remain confidential.
- Medical Journal Review: Upon request, all pertinent study data and information will be
  made available as supplemental information for journal editors and reviewers to evaluate
  and audit; eg, protocol and amendments and data tabulations. Arrangements will be
  made to maintain the confidentiality of such supplemental information. Arrangements
  will also be made to maintain the confidentiality of the identity of journal reviewers.
  Records will be maintained of which documents and datasets were reviewed.

#### 16. LIST OF REFERENCES

Brookhart MA. Counterpoint: The Treatment Decision Design. American Journal of Epidemiology. 2015;182:840–845.

Cameron, AC, Gelbach JB, Miller DL. Bootstrap-based improvements for inference with clustered errors. The Review of Economics and Statistics. 2008;90(3):414-427.

Chalasani NP, Hayashi PH, Bonkovsky HL, et al. ACG Clinical Guideline: the diagnosis and management of idiosyncratic drug-induced liver injury. Am J Gastroenterol. 2014 Jul;109(7):950-66.

Cole SR, Frangakis CE. The consistency statement in causal inference: a definition or an assumption? Epidemiology. 2009;20:3–5.

Corpechot C, Abenavoli L, Rabahi N, et al. Biochemical response to ursodeoxycholic acid and long-term prognosis in primary biliary cirrhosis. Hepatology. 2008;48(3):871-877.

Danaei G, Rodríguez LA, Cantero OF, et al. Observational data for comparative effectiveness research: an emulation of randomised trials of statins and primary prevention of coronary heart disease. Stat Methods Med Res. 2013;22:70–96.

Davison AC, Hinkley DV. Further Ideas in 'Bootstrap Methods and their Application'. Cambridge University Press 2013, pp. 70–135.

European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of cholestatic liver diseases. J Hepatol. 2009;51:237-267.

Fine JP, Gray RJ. A Proportional Hazards Model for the Subdistribution of a Competing Risk'. Journal of the American Statistical Association. 1999;94:496–509.

Glasheen WP, Cordier T, Gumpina R, et al. Charlson Comorbidity Index: ICD-9 Update and ICD-10 Translation. Am Health Drug Benefits. 2019;12:188-197.

Gran JM, Røysland K, Wolbers M, et al. A sequential Cox approach for estimating the causal effect of treatment in the presence of time-dependent confounding applied to data from the Swiss HIV Cohort Study. Stat Med. 2010;29:2757–2768.

Greenland S, Robins JM. Identifiability, exchangeability, and epidemiological confounding. Int J Epidemiol. 1986;15:413–419.

Hernán MA, Alonso A, Logan R, et al. Observational studies analyzed like randomized experiments: an application to postmenopausal hormone therapy and coronary heart disease. Epidemiology. 2008;19:766–779.

Hernán MA, Robins JM. Per-Protocol Analyses of Pragmatic Trials. N Engl J Med. 2017;377:1391–1398.

Kim WR, Lindor KD, Locke GR 3rd, et al. Epidemiology and natural history of primary biliary cirrhosis in a US community. Gastroenterology. 2000;119:1631-1636.

Kumagi T, Guindi M, Fischer SE, et al. Baseline ductopenia and treatment response predict long-term histological progression in primary biliary cirrhosis. Am J Gastroenterol. 2010;105(10):2186-2194.

Lash TL. Bias Analysis', in Lash, T. L. et al. (eds) Modern Epidemiology. 4th edn. Wolters Kluwer 2021, pp. 711–754.

Lindor KD, Gershwin ME, Poupon R, et al. Primary biliary cirrhosis: AASLD practice guidelines. Hepatology 2009;50:291-308.

Meyers RP, Shaheen AA, Fong A, et al. Validation of coding algorithms for the identification of patients with primary biliary cirrhosis using administrative data. Can J Gastroenterol. 2010:24:175-182.

Perez FM, Fisher H, Hiu S, et al. Patients with primary biliary cholangitis treated with long-term obeticholic acid in a trial-setting demonstrate better event-free survival than external controls from the GLOBAL PBC and UK-PBC study groups. Oral presentation at: American Association for the Study of Liver Disease; November, 2011; Anaheim, CA.

Pearl J. On the consistency rule in causal inference: axiom, definition, assumption, or theorem? Epidemiology. 2010;21:872–875.

Petersen ML, Porter KE, Gruber S, et al. Diagnosing and responding to violations in the positivity assumption. Stat Methods Med Res. 2012;21:31–54.

Sarvet AL, Wanis KN, Stensrud MJ, et al. A Graphical Description of Partial Exchangeability. Epidemiology. 2020; 31:365–368.

Sato T, Matsuyama Y. Marginal structural models as a tool for standardization. Epidemiology. 2003;14:680–686.

Schoenfeld DA. Sample-size formula for the proportional-hazards regression model. Biometrics. 1983;39(2):499-503.

Shook-Sa BE, Hudgens MG. Power and sample size for observational studies of point exposure effects [published online ahead of print, 2020 Nov 23]. Biometrics. 2020;10.1111/biom.13405. doi:10.1111/biom.13405.

US Food and Drug Administration. Framework for FDA's Real-World Evidence Program. December 2018: US Department of Health & Human Services; https://www.fda.gov/media/120060/download.

US Food and Drug Administration. Real-World Data: Assessing Electronic Health Records and Medical Claims Data To Support Regulatory Decision Making for Drug and Biological Products. Guidance for Industry. September 2021: US Department of Health & Human Services; https://www.fda.gov/media/152503/download

VanderWeele TJ. Concerning the consistency assumption in causal inference. Epidemiology. 2009;20:880–883.

Westreich D, Cole SR. Invited commentary: positivity in practice. Am J Epidemiol. 2010;171:674–681.

# APPENDIX A. LIST OF INCLUSION, EXCLUSION AND COVARIATE CODES

# INCLUSION/EXCLUSION CRITERIA CODES

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| Inclusion c | Inclusion criteria | |
| K74.3 | ICD10 | Primary biliary cholangitis |
| 571.6 | ICD9 | Biliary cirrhosis (for rule-out in the baseline period) |
| <b>Exclusion</b> c | riteria | |
| 0FY00Z1 | ICD10 pcs | Transplantation of liver, syngeneic, open approach |
| 0FY00Z0 | ICD10 pcs | Transplantation of Liver, Allogeneic, Open Approach |
| 47135 | HCPCS/<br>CPT-4 | Liver allotransplantation; orthotopic; partial or whole, from cadaver or living donor, any age |
| B17.10 | ICD10 | Acute hepatitis C without hepatic coma |
| B17.11 | ICD10 | Acute hepatitis C with hepatic coma |
| 070.41 | ICD9 | Acute hepatitis C with hepatic coma |
| 070.51 | ICD9 | Acute hepatitis C without mention of hepatic coma |
| B18.2 | ICD10 | Chronic viral hepatitis C |
| 070.44 | ICD9 | Chronic hepatitis C with hepatic coma |
| 070.54 | ICD9 | Chronic hepatitis C without mention of hepatic coma |
| 070.70 | ICD9 | Unspecified viral hepatitis C without hepatic coma |
| 070.71 | ICD9 | Unspecified viral hepatitis C with hepatic coma |
| B16.0 | ICD10 | Acute hepatitis B with delta-agent with hepatic coma |
| B16.1 | ICD10 | Acute hepatitis B with delta-agent without hepatic coma |
| B16.2 | ICD10 | Acute hepatitis B without delta-agent with hepatic coma |
| B16.9 | ICD10 | Acute hepatitis B without delta-agent and without hepatic coma |
| B17.0 | ICD10 | Acute delta-(super) infection of hepatitis B carrier |
| 070.20 | ICD9 | Viral hepatitis B with hepatic coma, acute or unspecified, without mention of hepatitis delta |
| 070.21 | ICD9 | Viral hepatitis B with hepatic coma, acute or unspecified, with hepatitis delta |
| 070.30 | ICD9 | Viral hepatitis B without mention of hepatic coma, acute or unspecified, without mention of hepatitis delta |
| 070.31 | ICD9 | Viral hepatitis B without mention of hepatic coma, acute or unspecified, with hepatitis delta |
| B18.0 | ICD10 | Chronic viral hepatitis B with delta-agent |
| B18.1 | ICD10 | Chronic viral hepatitis B without delta-agent |
| 070.23 | ICD9 | Chronic viral hepatitis B with hepatic coma with hepatitis delta |
| 070.22 | ICD9 | Chronic viral hepatitis B with hepatic coma without hepatitis delta |
| 070.33 | ICD9 | Chronic viral hepatitis B without mention of hepatic coma with hepatitis delta |
| 070.32 | ICD9 | Chronic viral hepatitis B without mention of hepatic coma without mention of hepatitis delta |
| K83.01 | ICD10 | Primary sclerosing cholangitis (2019-2021 only) |
| K70.0 | ICD10 | Alcoholic fatty liver |

| CODE | ТҮРЕ | DESCRIPTION |
|---|---|---|
| K70.10 | ICD10 | Alcoholic hepatitis without ascites |
| K70.11 | ICD10 | Alcoholic hepatitis with ascites |
| K70.2 | ICD10 | Alcoholic fibrosis and sclerosis of liver |
| K70.30 | ICD10 | Alcoholic cirrhosis of liver without ascites |
| K70.31 | ICD10 | Alcoholic cirrhosis of liver with ascites |
| K70.40 | ICD10 | Alcoholic hepatic failure without coma |
| K70.41 | ICD10 | Alcoholic hepatic failure with coma |
| K70.9 | ICD10 | Alcoholic liver disease, unspecified |
| 571.0 | ICD9 | Alcoholic fatty liver |
| 571.1 | ICD9 | Acute alcoholic hepatitis |
| 571.2 | ICD9 | Alcoholic cirrhosis of liver |
| 571.3 | ICD9 | Alcoholic liver damage, unspecified |
| C22.0 | ICD10 | Liver cell carcinoma |
| C22.8 | ICD10 | Malignant neoplasm of liver, primary, unspecified as to type |
| C22.9 | ICD10 | Malignant neoplasm of liver, not specified as primary or secondary |
| 155.0 | ICD9 | Malignant neoplasm of liver, primary |
| 155.2 | ICD9 | Malignant neoplasm of liver, not specified as primary or secondary |
| K76.7 | ICD10 | Hepatorenal syndrome |
| 572.4 | ICD9 | Hepatorenal syndrome |
| K76.81 | ICD10 | Hepatopulmonary syndrome |
| 573.5 | ICD9 | Hepatopulmonary syndrome |
| I27.21 | ICD10 | Secondary pulmonary arterial hypertension |
| K75.81 | ICD10 | Nonalcoholic steatohepatitis |
| 571.8 | ICD9 | Other chronic nonalcoholic liver disease |
| C00 | ICD10 | Malignant neoplasm of lip |
| C02 | ICD10 | Malignant neoplasm of other and unspecified parts of tongue |
| C03 | ICD10 | Malignant neoplasm of gum |
| C04 | ICD10 | Malignant neoplasm of floor of mouth |
| C05 | ICD10 | Malignant neoplasm of palate |
| C06 | ICD10 | Malignant neoplasm of other and unspecified parts of mouth |
| C08 | ICD10 | Malignant neoplasm of other and unspecified major salivary glands |
| C09 | ICD10 | Malignant neoplasm of tonsil |
| C10 | ICD10 | Malignant neoplasm of oropharynx |
| C11 | ICD10 | Malignant neoplasm of nasopharynx |
| C13 | ICD10 | Malignant neoplasm of hypopharynx |
| C14 | ICD10 | Malignant neoplasm of other and ill-defined sites in the lip, oral cavity & pharynx |
| C15 | ICD10 | Malignant neoplasm of esophagus |
| C16 | ICD10 | Malignant neoplasm of stomach |
| C17 | ICD10 | Malignant neoplasm of small intestine |
| C18 | ICD10 | Malignant neoplasm of colon |
| C21 | ICD10 | Malignant neoplasm of anus and anal canal |

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| C22 | ICD10 | Malignant neoplasm of liver and intrahepatic bile ducts |
| C24 | ICD10 | Malignant neoplasm of other and unspecified parts of biliary tract |
| C25 | ICD10 | Malignant neoplasm of pancreas |
| C26 | ICD10 | Malignant neoplasm of other and ill-defined digestive organs |
| C30 | ICD10 | Malignant neoplasm of nasal cavity and middle ear |
| C31 | ICD10 | Malignant neoplasm of accessory sinuses |
| C32 | ICD10 | Malignant neoplasm of larynx |
| C34 | ICD10 | Malignant neoplasm of bronchus and lung |
| C38 | ICD10 | Malignant neoplasm of heart, mediastinum and pleura |
| C39 | ICD10 | Malignant neoplasm of other and ill-defined sites in the respiratory system and intrathoracic organs |
| C40 | ICD10 | Malignant neoplasm of bone and articular cartilage of limbs |
| C41 | ICD10 | Malignant neoplasm of bone and articular cartilage of other and unspecified sites |
| C47 | ICD10 | Malignant neoplasm of peripheral nerves and autonomic nervous system |
| C48 | ICD10 | Malignant neoplasm of retroperitoneum and peritoneum |
| C49 | ICD10 | Malignant neoplasm of other connective and soft tissue |
| C50 | ICD10 | Malignant neoplasm of breast |
| C51 | ICD10 | Malignant neoplasm of vulva |
| C53 | ICD10 | Malignant neoplasm of cervix uteri |
| C54 | ICD10 | Malignant neoplasm of corpus uteri |
| C56 | ICD10 | Malignant neoplasm of ovary |
| C57 | ICD10 | Malignant neoplasm of other and unspecified female genital organs |
| C60 | ICD10 | Malignant neoplasm of penis |
| C62 | ICD10 | Malignant neoplasm of testis |
| C63 | ICD10 | Malignant neoplasm of other and unspecified male genital organs |
| C64 | ICD10 | Malignant neoplasm of kidney, except renal pelvis |
| C65 | ICD10 | Malignant neoplasm of renal pelvis |
| C66 | ICD10 | Malignant neoplasm of ureter |
| C67 | ICD10 | Malignant neoplasm of bladder |
| C68 | ICD10 | Malignant neoplasm of other and unspecified urinary organs |
| C69 | ICD10 | Malignant neoplasm of eye and adnexa |
| C70 | ICD10 | Malignant neoplasm of meninges |
| C71 | ICD10 | Malignant neoplasm of brain |
| C72 | ICD10 | Malignant neoplasm of spinal cord, cranial nerves and other parts of central nervous system |
| C74 | ICD10 | Malignant neoplasm of adrenal gland |
| C75 | ICD10 | Malignant neoplasm of other endocrine glands and related structures |
| C76 | ICD10 | Malignant neoplasm of other and ill-defined sites |
| C77 | ICD10 | Secondary and unspecified malignant neoplasm of lymph nodes |
| C78 | ICD10 | Secondary malignant neoplasm of respiratory and digestive organs |
| C79 | ICD10 | Secondary malignant neoplasm of other and unspecified sites |

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| C80 | ICD10 | Malignant neoplasm without specification of site |
| 140 | ICD9 | Malignant neoplasm of lip |
| 141 | ICD9 | Malignant neoplasm of tongue |
| 142 | ICD9 | Malignant neoplasm of major salivary glands |
| 143 | ICD9 | Malignant neoplasm of gum |
| 144 | ICD9 | Malignant neoplasm of floor of mouth |
| 145 | ICD9 | Malignant neoplasm of other and unspecified parts of mouth |
| 146 | ICD9 | Malignant neoplasm of oropharynx |
| 147 | ICD9 | Malignant neoplasm of nasopharynx |
| 148 | ICD9 | Malignant neoplasm of hypopharynx |
| 149 | ICD9 | Malignant neoplasm of other and ill-defined sites within the lip, oral cavity, and pharynx |
| 150 | ICD9 | Malignant neoplasm of esophagus |
| 151 | ICD9 | Malignant neoplasm of stomach |
| 152 | ICD9 | Malignant neoplasm of small intestine, including duodenum |
| 153 | ICD9 | Malignant neoplasm of colon |
| 154 | ICD9 | Malignant neoplasm of rectum, rectosigmoid junction, and anus |
| 155 | ICD9 | Malignant neoplasm of liver and intrahepatic bile ducts |
| 156 | ICD9 | Malignant neoplasm of gallbladder and extrahepatic bile ducts |
| 157 | ICD9 | Malignant neoplasm of pancreas |
| 158 | ICD9 | Malignant neoplasm of retroperitoneum and peritoneum |
| 159 | ICD9 | Malignant neoplasm of other and ill-defined sites within the digestive organs and peritoneum |
| 160 | ICD9 | Malignant neoplasm of nasal cavities, middle ear, and accessory sinuses |
| 161 | ICD9 | Malignant neoplasm of larynx |
| 162 | ICD9 | Malignant neoplasm of trachea, bronchus, and lung |
| 163 | ICD9 | Malignant neoplasm of pleura |
| 164 | ICD9 | Malignant neoplasm of thymus, heart, and mediastinum |
| 165 | ICD9 | Malignant neoplasm of other and ill-defined sites within the respiratory system and intrathoracic organs |
| 170 | ICD9 | Malignant neoplasm of bone and articular cartilage |
| 171 | ICD9 | Malignant neoplasm of connective and other soft tissue |
| 174 | ICD9 | Malignant neoplasm of female breast |
| 175 | ICD9 | Malignant neoplasm of male breast |
| 180 | ICD9 | Malignant neoplasm of cervix uteri |
| 182 | ICD9 | Malignant neoplasm of body of uterus |
| 183 | ICD9 | Malignant neoplasm of ovary and other uterine adnexa |
| 184 | ICD9 | Malignant neoplasm of other and unspecified female genital organs |
| 186 | ICD9 | Malignant neoplasm of testis |
| 187 | ICD9 | Malignant neoplasm of penis and other male genital organs |
| 188 | ICD9 | Malignant neoplasm of bladder |

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| 189 | ICD9 | Malignant neoplasm of kidney and other and unspecified urinary organs |
| 190 | ICD9 | Malignant neoplasm of eye |
| 191 | ICD9 | Malignant neoplasm of brain |
| 192 | ICD9 | Malignant neoplasm of other and unspecified parts of nervous system |
| 194 | ICD9 | Malignant neoplasm of other endocrine glands and related structures |
| 195 | ICD9 | Malignant neoplasm of other and ill-defined sites |
| 196 | ICD9 | Secondary and unspecified malignant neoplasm of lymph nodes |
| 197 | ICD9 | Secondary malignant neoplasm of respiratory and digestive systems |
| 198 | ICD9 | Secondary malignant neoplasm of other specified sites |
| 199 | ICD9 | Malignant neoplasm without specification of site |
| B20 | ICD10 | Human immunodeficiency virus infection |
| B21 | ICD10 | Human immunodeficiency virus [HIV] disease resulting in malignant neoplasms |
| B22 | ICD10 | Human immunodeficiency virus [HIV] disease resulting in other specified diseases |
| 042 | ICD9 | Human immunodeficiency virus [HIV] infection |
| M88.0 | ICD10 | Osteitis deformans of skull |
| M88.1 | ICD10 | Osteitis deformans of vertebrae |
| M88.811 | ICD10 | Osteitis deformans of right shoulder |
| M88.812 | ICD10 | Osteitis deformans of left shoulder |
| M88.819 | ICD10 | Osteitis deformans of unspecified shoulder |
| M88.821 | ICD10 | Osteitis deformans of right upper arm |
| M88.822 | ICD10 | Osteitis deformans of left upper arm |
| M88.829 | ICD10 | Osteitis deformans of unspecified upper arm |
| M88.831 | ICD10 | Osteitis deformans of right forearm |
| M88.832 | ICD10 | Osteitis deformans of left forearm |
| M88.839 | ICD10 | Osteitis deformans of unspecified forearm |
| M88.841 | ICD10 | Osteitis deformans of right hand |
| M88.842 | ICD10 | Osteitis deformans of left hand |
| M88.849 | ICD10 | Osteitis deformans of unspecified hand |
| M88.851 | ICD10 | Osteitis deformans of right thigh |
| M88.852 | ICD10 | Osteitis deformans of left thigh |
| M88.859 | ICD10 | Osteitis deformans of unspecified thigh |
| M88.861 | ICD10 | Osteitis deformans of right lower leg |
| M88.862 | ICD10 | Osteitis deformans of left lower leg |
| M88.869 | ICD10 | Osteitis deformans of unspecified lower leg |
| M88.871 | ICD10 | Osteitis deformans of right ankle and foot |
| M88.872 | ICD10 | Osteitis deformans of left ankle and foot |
| M88.879 | ICD10 | Osteitis deformans of unspecified ankle and foot |
| M88.88 | ICD10 | Osteitis deformans of other bones |
| M88.89 | ICD10 | Osteitis deformans of multiple sites |
| M88.9 | ICD10 | Osteitis deformans of unspecified bone |
| 731.0 | ICD9 | Osteitis deformans without mention of bone tumor |

Version 1.0: 24Jan2022 Page 56

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| S02 | ICD10 | Fracture of skull and facial bones |
| S12 | ICD10 | Fracture of cervical vertebra and other parts of neck |
| S22 | ICD10 | Fracture of rib(s), sternum and thoracic spine |
| S32 | ICD10 | Fracture of lumbar spine and pelvis |
| S42 | ICD10 | Fracture of shoulder and upper arm |
| S52 | ICD10 | Fracture of forearm |
| S62 | ICD10 | Fracture at wrist and hand level |
| S72 | ICD10 | Fracture of femur |
| S82 | ICD10 | Fracture of lower leg, including ankle |
| S92 | ICD10 | Fracture of foot and toe, except ankle |
| 800 | ICD9 | Fracture of vault of skull |
| 801 | ICD9 | Fracture of base of skull |
| 802 | ICD9 | Fracture of face bones |
| 803 | ICD9 | Other and unqualified skull fractures |
| 804 | ICD9 | Multiple fractures involving skull or face with other bones |
| 805 | ICD9 | Fracture of vertebral column without mention of spinal cord injury |
| 806 | ICD9 | Fracture of vertebral column with spinal cord injury |
| 807 | ICD9 | Fracture of rib(s) sternum larynx and trachea |
| 808 | ICD9 | Fracture of pelvis |
| 809 | ICD9 | Ill-defined fractures of bones of trunk |
| 810 | ICD9 | Fracture of clavicle |
| 811 | ICD9 | Fracture of scapula |
| 812 | ICD9 | Fracture of humerus |
| 813 | ICD9 | Fracture of radius and ulna |
| 814 | ICD9 | Fracture of carpal bone(s) |
| 815 | ICD9 | Fracture of metacarpal bone(s) |
| 816 | ICD9 | Fracture of one or more phalanges of hand |
| 817 | ICD9 | Multiple fractures of hand bones |
| 818 | ICD9 | Ill-defined fractures of upper limb |
| 819 | ICD9 | Multiple fractures involving both upper limbs and upper limb with rib(s) and sternum |
| 820 | ICD9 | Fracture of neck of femur |
| 821 | ICD9 | Fracture of other and unspecified parts of femur |
| 822 | ICD9 | Fracture of patella |
| 823 | ICD9 | Fracture of tibia and fibula |
| 824 | ICD9 | Fracture of ankle |
| 825 | ICD9 | Fracture of one or more tarsal and metatarsal bones |
| 826 | ICD9 | Fracture of one or more phalanges of foot |
| 827 | ICD9 | Other multiple and ill-defined fractures of lower limb |
| 828 | ICD9 | Multiple fractures involving both lower limbs lower with upper limb and lower limb(s) with rib(s) and sternum |
| 829 | ICD9 | Fracture of unspecified bones |

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| I85.01 | ICD10 | Esophageal varices with bleeding |
| I85.11 | ICD10 | Secondary esophageal varices with bleeding |
| 456.0 | ICD9 | Esophageal varices with bleeding |
| K70.11 | ICD10 | Alcoholic hepatitis with ascites |
| K70.31 | ICD10 | Alcoholic cirrhosis of liver with ascites |
| K71.51 | ICD10 | Toxic liver disease with chronic active hepatitis with ascites |
| R18.0 | ICD10 | Malignant ascites |
| R18.8 | ICD10 | Other ascites |
| 571.2 | ICD9 | Alcoholic cirrhosis of liver |
| 789.51 | ICD9 | Malignant ascites |
| 789.59 | ICD9 | Other ascites |
| J94.8 | ICD10 | Other specified pleural conditions |
| 511.8 | ICD9 | Other specified forms of pleural effusion, except tuberculous |
| 567.23 | ICD9 | Spontaneous bacterial peritonitis |
| K65.2 | ICD10 | Spontaneous bacterial peritonitis |
| B15.0 | ICD10 | Hepatitis A with hepatic coma |
| B16.0 | ICD10 | Acute hepatitis B with delta-agent with hepatic coma |
| B16.2 | ICD10 | Acute hepatitis B without delta-agent with hepatic coma |
| B17.11 | ICD10 | Acute hepatitis C with hepatic coma |
| B19.0 | ICD10 | Unspecified viral hepatitis with hepatic coma |
| B19.11 | ICD10 | Unspecified viral hepatitis B with hepatic coma |
| B19.21 | ICD10 | Unspecified viral hepatitis C with hepatic coma |
| K70.41 | ICD10 | Alcoholic hepatic failure with coma |
| K72.11 | ICD10 | Chronic hepatic failure with coma |
| K71.11 | ICD10 | Toxic liver disease with hepatic necrosis, with coma |
| K72.01 | ICD10 | Acute and subacute hepatic failure with coma |
| K72.91 | ICD10 | Hepatic failure, unspecified with coma |
| 572.2 | ICD9 | Hepatic encephalopathy |
| 070.0 | ICD9 | Viral hepatitis A with hepatic coma |
| 070.21 | ICD9 | Viral hepatitis B with hepatic coma, acute or unspecified, with hepatitis delta |
| 070.20 | ICD9 | Viral hepatitis B with hepatic coma, acute or unspecified, without mention of hepatitis delta |
| 070.2 | ICD9 | Viral hepatitis b with hepatic coma |
| 070.6 | ICD9 | Unspecified viral hepatitis with hepatic coma |
| 070.4 | ICD9 | Other specified viral hepatitis with hepatic coma |
| 070.41 | ICD9 | Acute hepatitis C with hepatic coma |
| 070.6 | ICD9 | Unspecified viral hepatitis with hepatic coma |
| 070.71 | ICD9 | Unspecified viral hepatitis C with hepatic coma |
| Z48.23 | ICD10 | Encounter for aftercare following liver transplant |
| V42.7 | ICD9 | Liver transplant status |
| T86.40 | ICD10 | Unspecified complication of liver transplant |
| T86.41 | ICD10 | Liver transplant rejection |

| CODE | ТҮРЕ | DESCRIPTION |
|--------|-------|-----------------------------------------|
| T86.42 | ICD10 | Liver transplant failure |
| T86.43 | ICD10 | Liver transplant infection |
| T86.49 | ICD10 | Other complications of liver transplant |
| 996.82 | ICD9 | Complications of transplanted liver |

# COVARIATE CODES (INLCUDING CHARLESON COMORBIDITY INDEX

| | | DESCRIPTION |
|---|---|---|
| CODE | TYPE | DESCRIPTION |
| K76.6 | ICD10 | Portal hypertension |
| 572.3 | ICD9 | Portal hypertension |
| I86.4 | ICD10 | Gastric varices |
| 456.8 | ICD9 | Varices of other sites (non-specific) |
| I85.00 | ICD10 | Esophageal varices without bleeding |
| I85.10 | ICD10 | Secondary esophageal varices without bleeding |
| 456.1 | ICD9 | Esophageal varices without mention of bleeding |
| 456.21 | ICD9 | Esophageal varices in diseases classified elsewhere, without mention of bleeding |
| K74.5 | ICD10 | Biliary cirrhosis, unspecified |
| K74.60 | ICD10 | Unspecified cirrhosis of liver |
| K74.69 | ICD10 | Other cirrhosis of liver |
| 571.5 | ICD9 | Cirrhosis of liver without mention of alcohol |
| I21 | ICD10 | Acute myocardial infarction |
| I22 | ICD10 | Subsequent ST elevation and non-ST elevation myocardial infarction |
| I25.2 | ICD10 | Old myocardial infarction |
| 410 | ICD9 | Acute myocardial infarction |
| 412 | ICD9 | Old myocardial infarction |
| I11.0 | ICD10 | Hypertensive heart disease with heart failure |
| I13.0 | ICD10 | Hypertensive heart and chronic kidney disease with heart failure and stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease |
| I13.2 | ICD10 | Hypertensive heart and chronic kidney disease with heart failure and with stage 5 chronic kidney disease, or end stage renal disease |
| I25.5 | ICD10 | Ischemic cardiomyopathy |
| I42.0 | ICD10 | Cardiomyopathy |
| I42.5 | ICD10 | Other restrictive cardiomyopathy |
| I42.6 | ICD10 | Alcoholic cardiomyopathy |
| I42.7 | ICD10 | Cardiomyopathy due to drug and external agent |
| I42.8 | ICD10 | Other cardiomyopathies |
| I42.9 | ICD10 | Cardiomyopathy, unspecified |
| I43 | ICD10 | Cardiomyopathy in diseases classified elsewhere |
| I50 | ICD10 | Heart failure |
| P29.0 | ICD10 | Neonatal cardiac failure |
| 398.91 | ICD9 | Rheumatic heart failure (congestive) |
| 402.01 | ICD9 | Malignant hypertensive heart disease with heart failure |
| 402.11 | ICD9 | Benign hypertensive heart disease with heart failure |
| 402.91 | ICD9 | Unspecified hypertensive disease with heart failure |
| 404.01 | ICD9 | Hypertensive heart and chronic kidney disease with heart failure and stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease. |
| 404.03 | ICD9 | Hypertensive heart and chronic kidney disease, malignant, with heart failure and with chronic kidney disease stage V or end stage renal disease |

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| 404.11 | ICD9 | Hypertensive heart and chronic kidney disease, benign, with heart failure and with chronic kidney disease stage I through stage IV, or unspecified |
| 404.13 | ICD9 | Hypertensive heart and chronic kidney disease, benign, with heart failure and chronic kidney disease stage V or end stage renal disease |
| 404.91 | ICD9 | Hypertensive heart and chronic kidney disease, unspecified, with heart failure and with chronic kidney disease stage I through stage IV, or unspecified |
| 404.93 | ICD9 | Hypertensive heart and chronic kidney disease, unspecified, with heart failure and chronic kidney disease stage V or end stage renal disease |
| 425.4 | ICD9 | Other primary cardiomyopathies |
| 425.5 | ICD9 | Alcoholic cardiomyopathy |
| 425.6 | ICD9 | Cardiomyopathy in Chagas disease |
| 425.7 | ICD9 | Nutritional and metabolic cardiomyopathy |
| 425.8 | ICD9 | Cardiomyopathy in other disease classified elsewhere |
| 425.9 | ICD9 | Secondary cardiomyopathy |
| 428 | ICD9 | unspecified, Heart failure |
| I70 | ICD10 | Atherosclerosis |
| I71 | ICD10 | Aortic aneurysm and dissection |
| I73.1 | ICD10 | Thromboangiitis obliterans [Buerger's disease] |
| I73.8 | ICD10 | Other specified peripheral vascular diseases |
| I73.9 | ICD10 | Peripheral vascular disease, unspecified |
| I77.1 | ICD10 | Stricture of artery |
| I79.0 | ICD10 | Aneurysm of aorta in diseases classified elsewhere |
| I79.1 | ICD10 | Aortitis in diseases classified elsewhere |
| I79.8 | ICD10 | Other disorders of arteries, arterioles, and capillaries in diseases classified elsewhere |
| K55.1 | ICD10 | Chronic vascular disorders of intestine |
| K55.8 | ICD10 | Other vascular disorders of intestine |
| K55.9 | ICD10 | Vascular disorder of intestine, unspecified |
| Z95.8 | ICD10 | Presence of other cardiac and vascular implants and grafts |
| Z95.9 | ICD10 | Presence of cardiac and vascular implant and graft, unspecified |
| 093.0 | ICD9 | Aneurysm of aorta, specified as syphilitic |
| 437.3 | ICD9 | Cerebral aneurysm, non-ruptured |
| 440 | ICD9 | Atherosclerosis |
| 441 | ICD9 | Aortic aneurysm and dissection |
| 443.1 | ICD9 | Thromboangiitis obliterans [Buerger's disease] |
| 443.2 | ICD9 | Other arterial dissection |
| 443.8 | ICD9 | Other specified peripheral vascular diseases |
| 443.9 | ICD9 | Peripheral vascular disease, unspecified |
| 447.1 | ICD9 | Stricture of artery |
| 557.1 | ICD9 | Chronic vascular insufficiency of intestine |
| 557.9 | ICD9 | Unspecified vascular insufficiency of intestine |
| V43.4* | ICD9 | Blood vessels replaced by other means |

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| G45 | ICD10 | Transient cerebral ischemic attacks and related syndromes |
| G46 | ICD10 | Vascular syndromes of brain in cerebrovascular diseases |
| H34.0 | ICD10 | Transient retinal artery occlusion |
| H34.1 | ICD10 | Central retinal artery occlusion |
| H34.2 | ICD10 | Other retinal artery occlusions |
| I60 | ICD10 | Non-traumatic subarachnoid hemorrhage |
| I61 | ICD10 | Non-traumatic intracerebral hemorrhage |
| I62 | ICD10 | Other and unspecified non-traumatic intracranial hemorrhage |
| I63 | ICD10 | Cerebral infarction |
| I64 | ICD10 | Stroke, not specified as hemorrhage or infarction |
| I65 | ICD10 | Occlusion and stenosis of precerebral arteries, not resulting in cerebral infarction |
| I66 | ICD10 | Occlusion and stenosis of cerebral arteries, not resulting in cerebral infarction |
| I67 | ICD10 | Other cerebrovascular diseases |
| I68 | ICD10 | Cerebrovascular disorders in diseases classified elsewhere |
| 362.34 | ICD9 | Transient retinal arterial occlusion |
| 430 | ICD9 | Subarachnoid hemorrhage |
| 431 | ICD9 | Intracerebral hemorrhage |
| 432 | ICD9 | Other and unspecified intracranial hemorrhage |
| 433 | ICD9 | Occlusion and stenosis of precerebral arteries |
| 434 | ICD9 | Occlusion of cerebral arteries |
| 435 | ICD9 | Transient cerebral ischemia |
| 436 | ICD9 | Acute, but ill-defined, cerebrovascular disease |
| 437 | ICD9 | Other and ill-defined cerebrovascular disease |
| 438 | ICD9 | Late effects of cerebrovascular disease |
| F01 | ICD10 | Vascular dementia |
| F02 | ICD10 | Dementia in other diseases classified elsewhere |
| F03 | ICD10 | Unspecified dementia |
| F04 | ICD10 | Amnestic disorder due to known physiological condition |
| F05 | ICD10 | Delirium due to known physiological condition |
| F06.1 | ICD10 | Catatonic disorder due to known physiological condition |
| F06.8 | ICD10 | Other specified mental disorders due to known physiological condition |
| G13.2 | ICD10 | Systemic atrophy primarily affecting the central nervous system in myxedema |
| G13.8 | ICD10 | Systemic atrophy primarily affecting central nervous system in other diseases classified elsewhere |
| G30 | ICD10 | Alzheimer's disease |
| G31.0 | ICD10 | Frontotemporal dementia |
| G31.1 | ICD10 | Senile degeneration of brain, not elsewhere classified |
| G31.2 | ICD10 | Degeneration of nervous system due to alcohol |
| G91.4 | ICD10 | Hydrocephalus in diseases classified elsewhere |
| G94 | ICD10 | Other disorders of brain in diseases classified elsewhere |
| R41.81 | ICD10 | Age-related cognitive decline |
| R54 | ICD10 | Age-related physical debility |

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| 290.0 | ICD9 | Senile dementia, uncomplicated |
| 290.1 | ICD9 | Presenile dementia |
| 290.2 | ICD9 | Senile dementia with delusional or depressive features |
| 290.3 | ICD9 | Senile dementia with delirium |
| 290.4 | ICD9 | Vascular dementia |
| 294.0 | ICD9 | Amnestic disorder in conditions classified elsewhere |
| 294.1 | ICD9 | Dementia in conditions classified elsewhere |
| 294.2 | ICD9 | mentia, unspecified |
| 294.8 | ICD9 | Other persistent mental disorders due to conditions classified elsewhere |
| 331.0 | ICD9 | Alzheimer's disease |
| 331.1 | ICD9 | Frontotemporal dementia |
| 331.2 | ICD9 | Senile degeneration of brain |
| 331.7 | ICD9 | Cerebral degeneration in diseases classified elsewhere |
| 797 | ICD9 | Senility without mention of psychosis |
| J40 | ICD10 | Bronchitis, not specified as acute or chronic |
| J41 | ICD10 | Simple and mucopurulent chronic bronchitis |
| J42 | ICD10 | Unspecified chronic bronchitis |
| J43 | ICD10 | Emphysema |
| J44 | ICD10 | Other chronic obstructive pulmonary disease |
| J45 | ICD10 | sthma |
| J46 | ICD10 | Status asthmaticus |
| J47 | ICD10 | Bronchiectasis |
| J60 | ICD10 | Coal worker's pneumoconiosis |
| J61 | ICD10 | Pneumoconiosis due to asbestos and other mineral fibers |
| J62 | ICD10 | Pneumoconiosis due to dust containing silica |
| J63 | ICD10 | Pneumoconiosis due to other inorganic dusts |
| J64 | ICD10 | Unspecified pneumoconiosis |
| J65 | ICD10 | Pneumoconiosis associated with tuberculosis |
| J66 | ICD10 | Airway disease due to specific organic dust |
| J67 | ICD10 | Hypersensitivity pneumonitis due to organic dust |
| J68.4 | ICD10 | Chronic respiratory conditions due to chemicals, gases, fumes and vapors |
| J70.1 | ICD10 | Chronic and other pulmonary manifestations due to radiation |
| J70.3 | ICD10 | Chronic drug-induced interstitial lung disorders |
| 490 | ICD9 | Bronchitis, not specified as acute or chronic |
| 491 | ICD9 | Chronic bronchitis |
| 492 | ICD9 | Emphysema |
| 493 | ICD9 | Asthma |
| 494 | ICD9 | Bronchiectasis |
| 495 | ICD9 | Extrinsic allergic alveolitis |
| 496 | ICD9 | Chronic airway obstruction, not elsewhere classified |
| 500 | ICD9 | Coal workers' pneumoconiosis |

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| 501 | ICD9 | Asbestosis |
| 502 | ICD9 | Pneumoconiosis due to other silica or silicates |
| 503 | ICD9 | Pneumoconiosis due to other inorganic dust |
| 504 | ICD9 | Pneumonopathy due to inhalation of other dust |
| 505 | ICD9 | Pneumoconiosis, unspecified |
| 506.4 | ICD9 | Chronic respiratory conditions due to fumes and vapors |
| 508.1 | ICD9 | Chronic and other pulmonary manifestations due to radiation |
| 508.8 | ICD9 | espiratory conditions due to other specified external agents |
| M05 | ICD10 | Rheumatoid arthritis with rheumatoid factor |
| M06 | ICD10 | Other rheumatoid arthritis |
| M31.5 | ICD10 | Giant cell arteritis with polymyalgia rheumatica |
| M32 | ICD10 | Systemic lupus erythematosus (SLE) |
| M33 | ICD10 | Dermatopolymyositis |
| M34 | ICD10 | Systemic sclerosis [scleroderma] |
| M35.1 | ICD10 | Other overlap syndromes |
| M35.3 | ICD10 | Polymyalgia rheumatica |
| M36.0 | ICD10 | Dermato(poly)myositis in neoplastic disease |
| 446.5 | ICD9 | Polyarteritis nodosa and allied conditions |
| 710.0 | ICD9 | ystemic lupus erythematosus |
| 710.1 | ICD9 | systemic sclerosis |
| 710.2 | ICD9 | icca syndrome |
| 710.3 | ICD9 | Dermatomyositis |
| 710.4 | ICD9 | olymyositis |
| 714.0 | ICD9 | Rheumatoid arthritis |
| 714.1 | ICD9 | Felty's syndrome |
| 714.2 | ICD9 | Other rheumatoid arthritis with visceral or systemic involvement |
| 714.8 | ICD9 | Other specified inflammatory polyarthropathies |
| 725 | ICD9 | Polymyalgia rheumatica |
| K25 | ICD10 | Gastric ulcer |
| K26 | ICD10 | Duodenal ulcer |
| K27 | ICD10 | Peptic ulcer, site unspecified |
| K28. | ICD10 | Gastrojejunal ulcer |
| 531 | ICD9 | Gastric ulcer |
| 532 | ICD9 | Duodenal ulcer |
| 533 | ICD9 | Peptic ulcer, site unspecified |
| 534 | ICD9 | Gastrojejunal ulcer |
| B18 | ICD10 | Chronic viral hepatitis |
| K70.0 | ICD10 | Alcoholic fatty liver |
| K70.1 | ICD10 | Alcoholic hepatitis |
| K70.2 | ICD10 | Alcoholic fibrosis and sclerosis of liver |
| K70.3 | ICD10 | Alcoholic cirrhosis of liver |

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| K70.9 | ICD10 | Alcoholic liver disease, unspecified |
| K71.3 | ICD10 | Toxic liver disease with chronic persistent hepatitis |
| K71.4 | ICD10 | Toxic liver disease with chronic lobular hepatitis |
| K71.5 | ICD10 | Toxic liver disease with chronic active hepatitis |
| K71.7 | ICD10 | Toxic liver disease with fibrosis and cirrhosis of liver |
| K73 | ICD10 | Chronic hepatitis, not elsewhere classified |
| K74 | ICD10 | Fibrosis and cirrhosis of liver |
| K76.0 | ICD10 | Fatty (change of) liver, not elsewhere classified |
| K76.2 | ICD10 | Central hemorrhagic necrosis of liver |
| K76.3 | ICD10 | Infarction of liver |
| K76.4 | ICD10 | Peliosis hepatis |
| K76.8 | ICD10 | Other specified diseases of liver |
| K76.9 | ICD10 | Liver disease, unspecified |
| Z94.4 | ICD10 | Liver transplant status |
| 070.22 | ICD9 | Chronic viral hepatitis B with hepatic coma without hepatitis delta |
| 070.23 | ICD9 | Chronic viral hepatitis B with hepatic coma with hepatitis delta |
| 070.32 | ICD9 | Chronic viral hepatitis B without mention of hepatic coma without mention of hepatitis delta |
| 070.33 | ICD9 | Chronic viral hepatitis B without mention of hepatic coma with hepatitis delta |
| 070.44 | ICD9 | Chronic hepatitis C with hepatic coma |
| 070.54 | ICD9 | Chronic hepatitis C without mention of hepatic coma |
| 070.6 | ICD9 | Unspecified viral hepatitis with hepatic coma |
| 070.9 | ICD9 | Unspecified viral hepatitis without mention of hepatic coma |
| 570 | ICD9 | Acute and subacute necrosis of liver |
| 571 | ICD9 | Chronic liver disease and cirrhosis |
| 573.3 | ICD9 | Hepatitis, unspecified |
| 573.4 | ICD9 | Hepatic infarction |
| 573.8 | ICD9 | Other specified disorders of liver |
| 573.9 | ICD9 | Unspecified disorder of liver |
| V42.7* | ICD9 | Liver replaced by transplant |
| E08 | ICD10 | Diabetes mellitus due to underlying condition |
| E09 | ICD10 | Drug or chemical induced diabetes mellitus |
| E10 | ICD10 | Type 1 diabetes mellitus |
| E11 | ICD10 | Type 2 diabetes mellitus |
| E13 | ICD10 | Other specified diabetes mellitus |
| 250.8 | ICD9 | Diabetes with other specified manifestations |
| 250.9 | ICD9 | Diabetes with unspecified complication |
| 249.0 | ICD9 | Secondary diabetes mellitus without mention of complication |
| 249.1 | ICD9 | Secondary diabetes mellitus with ketoacidosis |
| 249.2 | ICD9 | Secondary diabetes mellitus with hyperosmolarity |
| 249.3 | ICD9 | Secondary diabetes mellitus with other coma |
| 249.9 | ICD9 | Secondary diabetes mellitus with unspecified complication, no stated an uncontrolled, |

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| | | or unspecified |
| I12.9 | ICD10 | Hypertensive chronic kidney disease with stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease |
| I13.0 | ICD10 | Hypertensive heart and chronic kidney disease with heart failure and stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease |
| I13.10 | ICD10 | Hypertensive heart and CKD without heart failure with stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease |
| N03 | ICD10 | Chronic nephritic syndrome |
| N05 | ICD10 | Unspecified nephritic syndrome |
| N18.1 | ICD10 | Chronic kidney disease, Stage 1 |
| N18.2 | ICD10 | Chronic kidney disease, Stage 2 (mild) |
| N18.3 | ICD10 | Chronic kidney disease, Stage 3 (moderate) |
| N18.4 | ICD10 | Chronic kidney disease, Stage 4 (severe) |
| N18.9 | ICD10 | Chronic kidney disease, unspecified |
| Z94.0 | ICD10 | Kidney transplant status |
| 403.00 | ICD9 | Hypertensive chronic kidney disease, malignant, with chronic kidney disease stage I through stage IV, or unspecified |
| 403.10 | ICD9 | Hypertensive chronic kidney disease, malignant, with chronic kidney disease stage I through stage IV, or unspecified |
| 403.90 | ICD9 | Hypertensive chronic kidney disease, unspecified, with chronic kidney disease stage I through stage IV, or unspecified |
| 404.00 | ICD9 | Hypertensive heart and chronic kidney disease, malignant, without heart failure and with chronic kidney disease stage I through stage IV, or unspecified |
| 404.01 | ICD9 | Hypertensive heart and chronic kidney disease, malignant, with heart failure and with chronic kidney disease stage I through stage IV, or unspecified |
| 404.10 | ICD9 | Hypertensive heart and chronic kidney disease, benign, without heart failure and with chronic kidney disease stage I through stage IV, or unspecified |
| 404.11 | ICD9 | Hypertensive heart and chronic kidney disease, benign, with heart failure and with chronic kidney disease stage I through stage IV, or unspecified |
| 404.90 | ICD9 | Hypertensive heart and chronic kidney disease, unspecified, without heart failure and with chronic kidney disease stage I through stage IV, or unspecified |
| 404.91 | ICD9 | Hypertensive heart and chronic kidney disease, unspecified, with heart failure and with chronic kidney disease stage I through stage IV, or unspecified |
| 582 | ICD9 | Chronic glomerulonephritis |
| 583 | ICD9 | Nephritis/nephropathy |
| 585.1 | ICD9 | Chronic kidney disease, Stage I |
| 585.2 | ICD9 | Chronic kidney disease, Stage II (mild) |
| 585.3 | ICD9 | Chronic kidney disease, Stage III (moderate) |
| 585.4 | ICD9 | Chronic kidney disease, Stage IV (severe) |
| 585.9 | ICD9 | Chronic kidney disease, unspecified |

Page 66

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| V42.0 | ICD9 | Kidney replaced by transplant |
| E08 | ICD10 | Diabetes mellitus due to underlying condition |
| E09 | ICD10 | Drug or chemical induced diabetes mellitus |
| E10 | ICD10 | Type 1 diabetes mellitus |
| E11 | ICD10 | Type 2 diabetes mellitus |
| E13 | ICD10 | Other specified diabetes mellitus |
| 250.4 | ICD9 | Diabetes with renal manifestations |
| 250.5 | ICD9 | betes with ophthalmic complications |
| 250.6 | ICD9 | Diabetes with neurological manifestations |
| 250.7 | ICD9 | Diabetes with peripheral circulatory disorders |
| G04.1 | ICD10 | Tropical spastic paraplegia |
| G11.4 | ICD10 | Hereditary spastic paraplegia |
| G80.0 | ICD10 | Spastic quadriplegic cerebral palsy |
| G80.1 | ICD10 | Spastic diplegia cerebral palsy |
| G80.2 | ICD10 | Spastic hemiplegic cerebral palsy |
| G81 | ICD10 | Hemiplegia and hemiparesis |
| G82 | ICD10 | Paraplegia (paraparesis s) and quadriplegia |
| G83 | ICD10 | Other paralytic syndromes |
| 334.1 | ICD9 | Hereditary spastic paraplegia |
| 342 | ICD9 | Hemiplegia and hemiparesis |
| 343 | ICD9 | Infantile cerebral palsy |
| 344 | ICD9 | Other paralytic syndromes |
| I85.0 | ICD10 | Esophageal varices |
| I86.4 | ICD10 | Gastric varices |
| K70.4 | ICD10 | Alcoholic hepatic failure |
| K71.1 | ICD10 | Toxic liver disease with hepatic necrosis |
| K72.1 | ICD10 | Chronic hepatic failure |
| K72.9 | ICD10 | Hepatic failure, unspecified |
| K76.5 | ICD10 | Hepatic veno-occlusive disease |
| K76.6 | ICD10 | Portal hypertension |
| K76.7 | ICD10 | Hepatorenal syndrome |
| 456.0 | ICD9 | Esophageal varices with bleeding |
| 456.1 | ICD9 | Esophageal varices without mention of bleeding |
| 456.2 | ICD9 | Esophageal varices in diseases classified elsewhere |
| 572.2 | ICD9 | Hepatic encephalopathy |
| 572.3 | ICD9 | Portal hypertension |
| 572.4 | ICD9 | Hepatorenal syndrome |
| 572.8 | ICD9 | Other sequelae of chronic liver disease |
| I12.0 | ICD10 | Hypertensive chronic kidney disease with stage 5 chronic kidney disease or end stage renal disease |

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| I13.11 | ICD10 | Hypertensive heart and CKD without heart failure with stage 5 chronic kidney |
| 113.11 | ICDIO | disease, or end stage renal disease |
| I13.2 | ICD10 | Hypertensive heart and chronic kidney disease with heart failure and with stage 5 chronic kidney disease, or end stage renal disease |
| N18.5 | ICD10 | Chronic kidney disease, Stage 5 |
| N18.6 | ICD10 | End stage renal disease |
| N19 | ICD10 | Unspecified kidney failure |
| N25.0 | ICD10 | Renal osteodystrophy |
| Z49 | ICD10 | Encounter for care involving renal dialysis |
| Z99.2 | ICD10 | Dependence on renal dialysis |
| 403.01 | ICD9 | Hypertensive chronic kidney disease, malignant, with chronic kidney disease stage V or end stage renal disease |
| 403.11 | ICD9 | Hypertensive chronic kidney disease, benign, with chronic kidney disease stage V or end stage renal disease |
| 403.91 | ICD9 | Hypertensive chronic kidney disease, unspecified, with chronic kidney disease stage V or end stage renal disease |
| 404.02 | ICD9 | Hypertensive heart and chronic kidney disease, malignant, without heart failure and with chronic kidney disease stage V or end stage renal disease |
| 404.03 | ICD9 | Hypertensive heart and chronic kidney disease, malignant, with heart failure and with chronic kidney disease stage V or end stage renal disease |
| 404.12 | ICD9 | Hypertensive heart and chronic kidney disease, benign, without heart failure and with chronic kidney disease stage V or end stage renal disease |
| 404.13 | ICD9 | Hypertensive heart and chronic kidney disease, benign, with heart failure and chronic kidney disease stage V or end stage renal disease |
| 404.92 | ICD9 | Hypertensive heart and chronic kidney disease, unspecified, without heart failure and with chronic kidney disease stage V or end stage renal disease |
| 404.93 | ICD9 | Hypertensive heart and chronic kidney disease, unspecified, with heart failure and chronic kidney disease stage V or end stage renal disease |
| 585.5 | ICD9 | Chronic kidney disease, Stage V |
| 585.6 | ICD9 | End stage renal disease |
| 586 | ICD9 | Renal failure NOS |
| 588.0 | ICD9 | Renal osteodystrophy |
| V45.11 | ICD9 | Renal dialysis status |
| V45.12 | ICD9 | Noncompliance with renal dialysis |
| V56.0 | ICD9 | Encounter for extracorporeal dialysis |
| V56.1 | ICD9 | Fitting and adjustment of extracorporeal dialysis catheter |
| V56.2 | ICD9 | Fitting and adjustment of peritoneal dialysis catheter |
| V56.31 | ICD9 | Encounter for adequacy testing for hemodialysis |
| V56.32 | ICD9 | Encounter for adequacy testing for peritoneal dialysis |
| V56.8 | ICD9 | Encounter for other dialysis |

# BIOPSY AND IMAGING PROCEDURE CODES FOR CIRRHOSIS

| CODE | ТҮРЕ | DESCRIPTION |
|---|---|---|
| 47000 | HCPCS/CPT-4 | Biopsy of liver, needle |
| 47001 | HCPCS/CPT-4 | Biopsy of liver, needle |
| 47100 | HCPCS/CPT-4 | Excision procedures on the liver |
| 0FB00ZX | ICD10 pcs | Excision of Liver, Open Approach, Diagnostic |
| 0FB03ZX | ICD10 pcs | Excision of Liver, Percutaneous Approach, Diagnostic |
| 0FB04ZX | ICD10 pcs | Excision of Liver, Percutaneous Endoscopic Approach, Diagnostic |
| 0FB10ZX | ICD10 pcs | Excision of Right Lobe Liver, Open Approach, Diagnostic |
| 0FB13ZX | ICD10 pcs | Excision of Right Lobe Liver, Percutaneous Approach, Diagnostic |
| 0FB14ZX | ICD10 pcs | Excision of Right Lobe Liver, Percutaneous Endoscopic Approach, Diagnostic |
| 0FB20ZX | ICD10 pcs | Excision of Left Lobe Liver, Open Approach, Diagnostic |
| 0FB23ZX | ICD10 pcs | Excision of Left Lobe Liver, Percutaneous Approach, Diagnostic |
| 0FB24ZX | ICD10 pcs | Excision of Left Lobe Liver, Percutaneous Endoscopic Approach,<br>Diagnostic |
| 5012 | ICD9 pcs | Open liver biopsy |
| 5011 | ICD9 pcs | Closed liver biopsy (Closed (percutaneous) [needle] biopsy of liver) |
| 5014 | ICD9 pcs | Laparoscopic liver bx (Laparoscopic liver biopsy) |
| 91200 | HCPCS/CPT-4 | Nonimaging liver elastography |
| 76700 | HCPCS/CPT-4 | Complete ultrasound examination of the abdomen |
| 76705 | HCPCS/CPT-4 | Ultrasound, abdominal, real time with image documentation |
| BF45ZZZ | ICD10 pcs | Ultrasonography of Liver |
| BF46ZZZ | ICD10 pcs | Ultrasonography of Liver and Spleen |
| 8874 | ICD9 pcs | Dx ultrasound-digestive (Diagnostic ultrasound of digestive system) |
| 74181 | HCPCS/CPT-4 | MRI scan of abdomen |
| 74182 | HCPCS/CPT-4 | MRI scan of abdomen with contrast |
| 74183 | HCPCS/CPT-4 | MRI scan of abdomen before and after contrast |
| 74185 | HCPCS/CPT-4 | MRI scan of blood vessels of abdomen |
| BF35Y0Z | ICD10 pcs | Magnetic Resonance Imaging (MRI) of Liver using Other Contrast,<br>Unenhanced and Enhanced |
| BF35YZZ | ICD10 pcs | Magnetic Resonance Imaging (MRI) of Liver using Other Contrast |
| BF35ZZZ | ICD10 pcs | Magnetic Resonance Imaging (MRI) of Liver |
| 74150 | HCPCS/CPT-4 | CT imaging of the abdomen and pelvis |
| 74160 | HCPCS/CPT-4 | CT imaging of the abdomen |
| 74170 | HCPCS/CPT-4 | CT imaging of the abdomen with and without IV contrast |
| BF2500Z | ICD10 pcs | Computerized Tomography of Liver using High Osmolar Contrast,<br>Unenhanced and Enhanced |
| BF250ZZ | ICD10 pcs | Computerized Tomography of Liver using High Osmolar Contrast |
| BF2510Z | ICD10 pcs | Computerized Tomography of Liver using Low Osmolar Contrast, Unenhanced and Enhanced |
| BF251ZZ | ICD10 pcs | Computerized Tomography of Liver using Low Osmolar Contrast |
| BF25Y0Z | ICD10 pcs | Computerized Tomography of Liver using Other Contrast, Unenhanced and Enhanced |

| CODE | TYPE | DESCRIPTION |
|---|---|---|
| BF25YZZ | ICD10 pcs | Computerized Tomography of Liver using Other Contrast |
| BF25ZZZ | ICD10 pcs | Computerized Tomography of Liver |
| BF2600Z | ICD10 pcs | Computerized Tomography of Liver and Spleen using High Osmolar Contrast, Unenhanced and Enhanced |
| BF260ZZ | ICD10 pcs | Computerized Tomography of Liver and Spleen using High Osmolar Contrast |
| BF2610Z | ICD10 pcs | Computerized Tomography of Liver and Spleen using Low Osmolar Contrast, Unenhanced and Enhanced |
| BF261ZZ | ICD10 pcs | Computerized Tomography of Liver and Spleen using Low Osmolar Contrast |
| BF26Y0Z | ICD10 pcs | Computerized Tomography of Liver and Spleen using Other Contrast, Unenhanced and Enhanced |
| BF26YZZ | ICD10 pcs | Computerized Tomography of Liver and Spleen using Other Contrast |
| BF26ZZZ | ICD10 pcs | Computerized Tomography of Liver and Spleen |
| BF2C00Z | ICD10 pcs | Computerized Tomography of Hepatobiliary System, All using High Osmolar Contrast, Unenhanced and Enhanced |
| BF2C0ZZ | ICD10 pcs | Computerized Tomography of Hepatobiliary System, All using High<br>Osmolar Contrast |
| BF2C10Z | ICD10 pcs | Computerized Tomography of Hepatobiliary System, All using Low Osmolar Contrast, Unenhanced and Enhanced |
| BF2C1ZZ | ICD10 pcs | Computerized Tomography of Hepatobiliary System, All using Low Osmolar Contrast |
| BF2CY0Z | ICD10 pcs | Computerized Tomography of Hepatobiliary System, All using Other Contrast, Unenhanced and Enhanced |
| BF2CYZZ | ICD10 pcs | Computerized Tomography of Hepatobiliary System, All using Other Contrast |
| BF2CZZZ | ICD10 pcs | Computerized Tomography of Hepatobiliary System, All |
| BW2000Z | ICD10 pcs | Computerized Tomography of Abdomen using High Osmolar Contrast, Unenhanced and Enhanced |
| BW200ZZ | ICD10 pcs | Computerized Tomography of Abdomen using High Osmolar<br>Contrast |
| BW2010Z | ICD10 pcs | Computerized Tomography of Abdomen using Low Osmolar<br>Contrast, Unenhanced and Enhanced |
| BW201ZZ | ICD10 pcs | Computerized Tomography of Abdomen using Low Osmolar<br>Contrast |
| BW20Y0Z | ICD10 pcs | Computerized Tomography of Abdomen using Other Contrast,<br>Unenhanced and Enhanced |
| BW20YZZ | ICD10 pcs | Computerized Tomography of Abdomen using Other Contrast |
| BW20ZZZ | ICD10 pcs | Computerized Tomography of Abdomen |

# APPENDIX B. TABLE SHELLS

# Table 1A: Eligibility Criteria June 2015 to December 2021 (Komodo Health Only)

| | All Patients<br>N = XX |
|---|---|
| Eligibility Criteria | n (%) |
| All patients with PBC code | |
| PBC diagnosis | |
| 1 inpatient claim | |
| 2 outpatient claims | |
| 1 inpatient and/or 2 outpatient claims | |
| PBC Dx + Laboratory data | |
| ALP | |
| Bilirubin | |
| AST | |
| ALT | |
| ALP and Bilirubin and AST and ALT | |
| PBC Dx + Labs + Prescription record for UDCA | |
| PBC Dx + Labs + UDCA failure | |
| UDCA intolerant | |
| Inadequate UDCA response | |
| PBC Dx + Labs + UDCA failure + 12 months data before UDCA failure | |
| PBC Dx + Labs + UDCA failure + 12 months pre-index data + 12 months closed claims | |
| PBC Dx + Labs + UDCA failure + 12 months pre-index data + 12 months closed claims + OCA | |

Table 1B: Eligibility Criteria June 2015 to December 2021 (Global PBC Registry Only)

| | All Patients N = XX |
|---|---|
| Eligibility Criteria | n (%) |
| All patients with PBC diagnosis | |
| PBC Dx + Laboratory data | |
| ALP | |
| Bilirubin | |
| AST | |
| ALT | |
| ALP and Bilirubin and AST and ALT | |
| PBC Dx + Labs + Prescription record for UDCA | |
| PBC Dx + Labs + UDCA failure | |
| UDCA intolerant | |
| Inadequate UDCA response | |
| PBC Dx + Labs + UDCA failure + 12 months data before UDCA failure | |
| PBC Dx + Labs + UDCA failure + 12 months pre-index data + OCA | |

**Table 2:** Sex of All Eligible Patients by Year

| | | All Eligible Patients | | | | | |
|---|---|---|---|---|---|---|---|
| | 2016<br>N=X | 2017<br>N=X | 2018<br>N=X | 2019<br>N=X | 2020<br>N=X | 2021<br>N=X | Overall<br>N=X |
| Sex | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Female | | | | | | | |
| Male | | | | | | | |
| Missing | | | | | | | |

Table 3: Age of All Eligible Patients by Year

| | All Eligible Patients | | | | | | |
|---|---|---|---|---|---|---|---|
| | 2016 | 2017 | 2018 | 2019 | 2020 | 2021 | Overall |
| Age | N=X | N=X | N=X | N=X | N=X | N=X | N=X |
| Valid, n (%) | | | | | | | |
| Missing, n (%) | | | | | | | |
| Mean (SD) | | | | | | | |
| Skewness | | | | | | | |
| Median | | | | | | | |
| (Q1, Q3) | | | | | | | |
| Range | | | | | | | |

Table 4: Race of All Eligible Patients by Year\*

| | All Eligible Patients | | | | | | |
|---|---|---|---|---|---|---|---|
| | 2016<br>N=X | 2017<br>N=X | 2018<br>N=X | 2019<br>N=X | 2020<br>N=X | 2021<br>N=X | Overall<br>N=X |
| Race | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| White | | | | | | | |
| Black or African American | | | | | | | |
| Asian, Native Hawaiian or other Pacific Islander | | | | | | | |
| American Indian or Alaskan<br>Native | | | | | | | |
| Other | | | | | | | |
| Missing | | | | | | | |

<sup>\*</sup> Note that race is not systematically reported in either database, and thus is only available on a subset of patients.

**Table 5A:** Region by Year (Komodo Health Only)

| | All Eligible Patients | | | | | | |
|---|---|---|---|---|---|---|---|
| | 2016<br>N=X | 2017<br>N=X | 2018<br>N=X | 2019<br>N=X | 2020<br>N=X | 2021<br>N=X | Overall<br>N=X |
| Region | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Northeast | | | | | | | |
| Midwest | | | | | | | |
| West | | | | | | | |
| South | | | | | | | |
| Missing, n (%) | | | | | | | |
Table 5B: Patients by Country and by Year (Global PBC Registry Only)

| | All Eligible Patients | | | | | | |
|---|---|---|---|---|---|---|---|
| | 2016 | 2017 | 2018 | 2019 | 2020 | 2021 | Overall |
| | N=X | N=X | N=X | N=X | N=X | N=X | N=X |
| Country | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| The Netherlands | | | | | | | |
| UK | | | | | | | |
| Belgium | | | | | | | |
| Germany | | | | | | | |
| France | | | | | | | |
| Italy | | | | | | | |
| Spain | | | | | | | |
| Greece | | | | | | | |
| Canada | | | | | | | |
| USA | | | | | | | |
| Argentina | | | | | | | |
| Israel | | | | | | | |
| Japan | | | | | | | |
| China | | | | | | | |

 Table 6:
 Index Hepatic Laboratory Values by Year (TB, ALP, ALT, AST)

| | All Eligible Patients | | | | | | |
|---|---|---|---|---|---|---|---|
| Laboratory Value<br>Statistic | 2016<br>N pts=X<br>N index =X | 2017<br>N pts=X<br>N index =X | 2018<br>N pts=X<br>N index =X | 2019<br>N pts=X<br>N index =X | 2020<br>N pts=X<br>N index =X | 2021<br>N pts=X<br>N index =X | Overall N pts=X N index =X |
| ТВ | | | | | | | |
| Valid, n (%) | | | | | | | |
| Missing, n (%) | | | | | | | |
| Mean (SD) | | | | | | | |
| Skewness | | | | | | | |
| Median | | | | | | | |
| (Q1, Q3) | | | | | | | |
| Range | | | | | | | |
| ALP | | | | | | | |
| Valid, n (%) | | | | | | | |
| Missing, n (%) | | | | | | | |
| Mean (SD) | | | | | | | |
| Skewness | | | | | | | |
| Median | | | | | | | |
| (Q1, Q3) | | | | | | | |
| Range | | | | | | | |
| ALT | | | | | | | |
| Valid, n (%) | | | | | | | |
| Missing, n (%) | | | | | | | |
| Mean (SD) | | | | | | | |
| Skewness | | | | | | | |
| Median | | | | | | | |
| (Q1, Q3) | | | | | | | |
| Range | | | | | | | |
| AST | | | | | | | |
| Valid, n (%) | | | | | | | |
| Missing, n (%) | | | | | | | |
| Mean (SD) | | | | | | | |
| Skewness | | | | | | | |
| Median | | | | | | | |
| (Q1, Q3) | | | | | | | |
| Range | | | | | | | |

**Table 7:** Index Platelet Counts by Year

| | All Eligible Patients | | | | | | |
|---|---|---|---|---|---|---|---|
| Platelet counts | 2016<br>N pts=X<br>N index =X | 2017<br>N pts=X<br>N index =X | 2018<br>N pts=X<br>N index =X | 2019<br>N pts=X<br>N index =X | 2020<br>N pts=X<br>N index =X | 2021<br>N pts=X<br>N index =X | Overall<br>N pts=X<br>N index =X |
| Valid, n (%) | | | | | | | |
| Missing, n (%) | | | | | | | |
| Mean (SD) | | | | | | | |
| Skewness | | | | | | | |
| Median | | | | | | | |
| (Q1, Q3) | | | | | | | |
| Range | | | | | | | |

**Table 8:** On UDCA Treatment by Year

| | All Eligible Patients<br>N=X |
|-------------------|------------------------------|
| On UDCA treatment | n (%) |
| 2016 | |
| 2017 | |
| 2019 | |
| 2020 | |
| 2021 | |

**Table 9: UDCA Failure by Year** 

| | All Eligible Patients<br>N=X |
|--------------|------------------------------|
| UDCA failure | n (%) |
| 2016 | |
| 2017 | |
| 2019 | |
| 2020 | |
| 2021 | |

Table 10: Time (Months) Since First UDCA Failure Until the Index Date (inclusive) by Year

| | All Eligible Patients | | | | | | |
|---|---|---|---|---|---|---|---|
| Months since UDCA failure until index date | 2016<br>N=X | 2017<br>N=X | 2018<br>N=X | 2019<br>N=X | 2020<br>N=X | 2021<br>N=X | Overall<br>N=X |
| Valid, n (%) | | | | | | | |
| Missing, n (%) | | | | | | | |
| Mean (SD) | | | | | | | |
| Skewness | | | | | | | |
| Median | | | | | | | |
| (Q1, Q3) | | | | | | | |
| Range | | | | | | | |

Table 11: Clinical Evidence of Portal Hypertension (Platelets <150k; Non-Bleeding Varices; Platelets and/or Non-Bleeding Varices) by Year

| | All Eligible Patients<br>N=X |
|---|---|
| Clinical evidence of portal hypertension by year | n (%) |
| 2016 | |
| 2017 | |
| 2019 | |
| 2020 | |
| 2021 | |

Table 12: Cirrhosis by Year

| | All Eligible Patients<br>N=X |
|-------------------|------------------------------|
| Cirrhosis by year | n (%) |
| 2016 | |
| 2017 | |
| 2019 | |
| 2020 | |
| 2021 | |

Table 13: Charlson Comorbidity Index Score by Year

| | All Eligible Patients | | | | | | |
|---|---|---|---|---|---|---|---|
| Charlson Comorbidity<br>Index Score by year | 2016<br>N=X | 2017<br>N=X | 2018<br>N=X | 2019<br>N=X | 2020<br>N=X | 2021<br>N=X | Overall<br>N=X |
| Valid, n (%) | | | | | | | |
| Missing, n (%) | | | | | | | |
| Mean (SD) | | | | | | | |
| Skewness | | | | | | | |
| Median | | | | | | | |
| (Q1, Q3) | | | | | | | |
| Range | | | | | | | |

**Table 14:** Insurance Type at Index Date by Year (Komodo Health Only)

| | | All Eligible Patients | | | | | |
|---|---|---|---|---|---|---|---|
| Health Insurance Type on | 2016<br>N=X | 2017<br>N=X | 2018<br>N=X | 2019<br>N=X | 2020<br>N=X | 2021<br>N=X | Overall<br>N=X |
| the index date | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Commercial | | | | | | | |
| Self-insured/Exchanges | | | | | | | |
| Medicare | | | | | | | |
| Medicaid | | | | | | | |
| Dual eligible | | | | | | | |
| Other | | | | | | | |
| Missing | | | | | | | |

**Table 15:** Number of Index Dates by Year

| | Year | | | | | | |
|---|---|---|---|---|---|---|---|
| Patients | 2016 | 2017 | 2018 | 2019 | 2020 | 2021 | Overall |
| Statistic | N=X | N=X | N=X | N=X | N=X | N=X | N=X |
| All Eligible Patients | | | | | | | |
| Patients with index date | | | | | | | |
| # index dates/patient with index date | | | | | | | |
| Mean (SD) | | | | | | | |
| Skewness | | | | | | | |
| Median | | | | | | | |
| (Q1, Q3) | | | | | | | |
| Range | | | | | | | |
| Non-OCA | | | | | | | |
| Patients with index date | | | | | | | |
| # index dates/patient with index date | | | | | | | |
| Mean (SD) | | | | | | | |
| Skewness | | | | | | | |
| Median | | | | | | | |
| (Q1, Q3) | | | | | | | |
| Range | | | | | | | |
| OCA | | | | | | | |
| Patients with index date | | | | | | | |
| # index dates/patient with index date | | | | | | | |
| Mean (SD) | | | | | | | |
| Skewness | | | | | | | |
| Median | | | | | | | |
| (Q1, Q3) | | | | | | | |
| Range | | | | | | | |

**Table 16:** Sex of Patients by Group before and After Weighting

| | Before W | eighting | After Weighting | |
|---|---|---|---|---|
| | Non-OCA-treated OCA-treated I | | Non-OCA-treated | OCA-treated |
| | N patients = | N patients = | N patients = | N patients = |
| | N index dates = | N index dates = | N index dates = | N index dates = |
| Sex | n (%) | n (%) | n (%) | n (%) |
| Female | | | | |
| Male | | | | |

**Table 17:** Age of Patients by Group Before and After Weighting

| | Before W | eighting | After Weighting | |
|---|---|---|---|---|
| | Non-OCA-treated | on-OCA-treated OCA-treated | | OCA-treated |
| | N patients = | N patients = | N patients = | N patients = |
| Age | N index dates = | N index dates = | N index dates = | N index dates = |
| Mean (SD) | | | | |
| Skewness | | | | |
| Median | | | | |
| (Q1, Q3) | | | | |
| Range | | | | |

Table 18A: Region by Group Before and After Weighting (Komodo Health Only)

| | Before W | eighting | After Weighting | |
|---|---|---|---|---|
| | Non-OCA-treated | OCA-treated | Non-OCA-treated | OCA-treated |
| | N patients = | N patients = | N patients = | N patients = |
| | N index dates = | N index dates = | N index dates = | N index dates = |
| Region | n (%) | n (%) | n (%) | n (%) |
| Northeast | | | | |
| Midwest | | | | |
| West | | | | |
| South | | | | |
| Missing | | | | |

Table 18B: Country by Group Before and After Weighting (Global PBC Registry Only)

| | Before W | Veighting | After Weighting | |
|---|---|---|---|---|
| | Non-OCA-treated | OCA-treated | Non-OCA-treated | OCA-treated |
| | N patients = | N patients = | N patients = | N patients = |
| | N index dates = | N index dates = | N index dates = | N index dates = |
| Countries in<br>Global PBC | n (%) | n (%) | n (%) | n (%) |

Table 19: Hepatic Laboratory Values by Group (TB, ALP, ALT, AST) Before and After Weighting

| | Before W | eighting | After Weighting | |
|---|---|---|---|---|
| | Non-OCA-treated | OCA-treated | Non-OCA-treated | OCA-treated |
| Hepatic | N patients = | N patients = | N patients = | N patients = |
| Laboratory Value | N index dates = | N index dates = | N index dates = | N index dates = |
| Statistic<br>TB | N index dates = | N index dates = | N index dates = | N index dates = |
| n (%) | | | | |
| Mean (SD) | | | | |
| Skewness | | | | |
| Median | | | | |
| (Q1, Q3) | | | | |
| Range | | | | |
| ALP | | | | |
| n (%) | | | | |
| Mean (SD) | | | | |
| Skewness | | | | |
| Median | | | | |
| (Q1, Q3) | | | | |
| Range | | | | |
| ALT | | | | |
| n (%) | | | | |
| Mean (SD) | | | | |
| Skewness | | | | |
| Median | | | | |
| (Q1, Q3) | | | | |
| Range | | | | |
| AST | | | | |
| n (%) | | | | |
| Mean (SD) | | | | |
| Skewness | | | | |
| Median | | | | |
| (Q1, Q3) | | | | |
| Range | | | | |

**Table 20:** Platelet Counts by Group Before and After Weighting

| | Before Weighting | | After Weighting | |
|---|---|---|---|---|
| | Non-OCA-treated OCA-treated | | Non-OCA-treated | OCA-treated |
| | N patients = | N patients = | N patients = | N patients = |
| Platelet counts | N index dates = | N index dates = | N index dates = | N index dates = |
| n (%) | | | | |
| Mean (SD) | | | | |
| Skewness | | | | |
| Median | | | | |
| (Q1, Q3) | | | | |
| Range | | | | |

**Table 21:** Patients on UDCA Treatment by Group Before and After Weighting

| | Before W | Veighting | After Weighting | |
|---|---|---|---|---|
| | Non-OCA-treated OCA-treated I | | Non-OCA-treated | OCA-treated |
| | N patients = N patients = | | N patients = | N patients = |
| | N index dates = | N index dates = | N index dates = | N index dates = |
| UDCA Treatment | n (%) | n (%) | n (%) | n (%) |
| Yes | | | | |
| No | | - | | |

Table 22: Duration (Months) of Receiving UDCA by Group Before and After Weighting

| | Before Weighting | | After Weighting | |
|---|---|---|---|---|
| | Non-OCA-treated | Non-OCA-treated OCA-treated | | OCA-treated |
| Duration (in | N patients = | N patients = | N patients = | N patients = |
| months) of UDCA treatment | N index dates = N index dates = | | N index dates = | N index dates = |
| Mean (SD) | | | | |
| Skewness | | | | |
| Median | | | | |
| (Q1, Q3) | | | | |
| Range | | | | |

Table 23: Time (Months) from UDCA Failure Until the Index Date by Group Before and After Weighting

| | Before Weighting | | After Weighting | |
|---|---|---|---|---|
| | Non-OCA-treated | OCA-treated | Non-OCA-treated | OCA-treated |
| Time (in months) | N patients = | N patients = | N patients = | N patients = |
| from UDCA failure until the index date | N index dates = N index dates = | | N index dates = | N index dates = |
| Mean (SD) | | | | |
| Skewness | | | | |
| Median | | | | |
| (Q1, Q3) | | | | |
| Range | | | | |

Table 24: Clinical Evidence of Portal Hypertension (Platelets <150k; Non-Bleeding Varices; Platelets and/or Non-Bleeding Varices) by Group Before and After Weighting

| | Before W | eighting | After Weighting | |
|---|---|---|---|---|
| | Non-OCA-treated | OCA-treated | Non-OCA-treated | OCA-treated |
| | N patients = | N patients = | N patients = | N patients = |
| Clinical evidence<br>of portal<br>hypertension | N index dates = | N index dates = | N index dates = | N index dates = |
| | n (%) | n (%) | n (%) | n (%) |
| Yes | | | | |
| No | | | | |

**Table 25:** Cirrhosis by Group Before and After Weighting

| | Before W | eighting | After Weighting | |
|---|---|---|---|---|
| | Non-OCA-treated OCA-treated | | Non-OCA-treated | OCA-treated |
| | N patients = N patients = | | N patients = | N patients = |
| | N index dates = N index dates = | | N index dates = | N index dates = |
| Cirrhosis | n (%) | n (%) | n (%) | n (%) |
| Yes | | | | |
| No | | | | |

Table 26: Charlson Comorbidity Index Score by Group Before and After Weighting

| | Before Weighting | | | After Weighting | | | | |
|---|---|---|---|---|---|---|---|---|
| | Non-OC | A-treated | OCA- | treated | Non-OC. | A-treated | OCA-1 | treated |
| Charlson | N patients = N patients = N index date | | N pati | ients = | N pat | ients = | N pati | ients = |
| Comorbidity Index<br>Score | | | dates = | N index dates = | | N index dates = | | |
| Mean (SD) | | | | | | | | |
| Skewness | | | | | | | | |
| Median | | | | | | | | |
| (Q1, Q3) | | | | | | | | |
| Range | | | | | | | | |

Table 27: Insurance Type at Index Date by Group Before and After Weighting (Komodo Health Only)

| | Before W | eighting | After Weighting | |
|---|---|---|---|---|
| | Non-OCA-treated | OCA-treated | Non-OCA-treated | OCA-treated |
| | N patients = | N patients = | N patients = | N patients = |
| Ton one of a section | N index dates = | N index dates = | N index dates = | N index dates = |
| Insurance type at index date | n (%) | n (%) | n (%) | n (%) |
| Commercial | | | | |
| Medicare | | | | |
| Medicaid | | | | |
| Dual eligible | | | | |
| Other | | | | |
| Missing | | | | |

 Table 28:
 Logistic regression for Non-OCA vs OCA-treated

| Parameter | N | Estimate | SE |
|--------------------------------------|---|----------|----|
| Non-OCA | | | |
| OCA | | | |
| Gender | | | |
| Age | | | |
| Region/Country | | | |
| Time (in months) since PBC diagnosis | | | |
| Calendar year of PBC diagnosis | | | |
| Labs | | | |
| ALP | | | |
| Total bilirubin | | | |
| ALT | | | |
| AST | | | |
| UDCA duration | | | |
| Clinical evidence of portal HTN | | | |
| Cirrhosis | | | |
| Charlson Comorbidity Index Score | | | |
| Insurance type | | | |

**Table 29:** Distribution of Propensity Weights

| | Non-OCA-treated | OCA-treated |
|--------------------|-----------------|-----------------|
| | N patients = | N patients = |
| Propensity weights | N index dates = | N index dates = |
| Mean (SD) | | |
| Skewness | | |
| Median | | |
| (Q1, Q3) | | |
| Range | | |

Table 30: Standardized Differences of the Mean Before and After Weighting

| | Standardized Mean Difference | |
|---|---|---|
| Parameter | Unweighted | Weighted |
| Gender | | |
| Age | | |
| Region/Country | | |
| Time (in months) since PBC diagnosis | | |
| Calendar year of PBC diagnosis | | |
| ALP | | |
| Total bilirubin | | |
| ALT | | |
| AST | | |
| UDCA duration | | |
| Clinical evidence of portal HTN | | |
| Cirrhosis | | |
| Charlson Comorbidity Index Score | | |
| Insurance type | | |

Table 31: Results Unadjusted, Adjusted and Weighted Cox Regression on Time to Composite Event

| Parameter | n | HR | 95% CI | p-value |
|----------------------------------|---|----|--------|---------|
| Unique cases | | | | |
| Unique persons | | | | |
| Cases | | | | |
| Person trials | | | | |
| Unadjusted | | | | |
| Adjusted for baseline covariates | | | | |
| Weighted | | | | |

Figure 1: Adherence to OCA Treatment over Time



Figure 2A: Eligible Patients by Number of Trials



Figure 2B: Eligible Control Patients by Number of Trials



Figure 2C: Eligible OCA-treated Patients by Number of Trials



Figure 3A: Distribution of Propensity Scores: Unweighted



Figure 3B: Distribution of Propensity Scores: Weighted



Figure 4: Kaplan-Meier Survival Curve: Composite Event-free Survival by Treatment Arm

